CLINICAL TRIAL: NCT02491463
Title: A Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK Biologicals' RSV Investigational Vaccine Based on Viral Proteins Encoded by Chimpanzee-derived Adenovector (ChAd155-RSV) (GSK3389245A) in Healthy Adults
Brief Title: A Study to Assess the Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' RSV Investigational Vaccine (ChAd155-RSV) (GSK3389245A) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201974
Record Dates: First submitted 2015-06-29; First posted 2015-07-08 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Synctial Virus Infections
Keywords: Reactogenicity; Safety; Respiratory syncytial virus (RSV); Vaccine; Immunogenicity
MeSH Terms: interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- GSK3389245A_LD GROUP (Experimental): Subjects in this group will receive 2 doses, one month apart of the GSK3389245A vaccine low dose
  Interventions: Biological: GSK3389245A_LD GROUP
- GSK3389245A_HD GROUP (Experimental): Subjects in this group will receive 2 doses, one month apart, of the GSK3389245A vaccine high dose
  Interventions: Biological: GSK3389245A_HD GROUP
- Bexsero Group (Active Comparator): Subjects in this group will receive 2 doses, one month apart, of Bexsero
  Interventions: Biological: Bexsero
- Placebo Group (Placebo Comparator): Subjects in this group will receive 2 doses, one month apart, of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: GSK3389245A_LD GROUP — 2 doses administered intramuscularly at Day 0 and Day 30 in the deltoid region of the non-dominant arm
  Arms: GSK3389245A_LD GROUP
Biological: GSK3389245A_HD GROUP — 2 doses administered intramuscularly at Day 0 and Day 30 in the deltoid region of the non-dominant arm
  Arms: GSK3389245A_HD GROUP
Biological: Bexsero — 2 doses administered intramuscularly at Day 0 and Day 30 in the deltoid region of the non-dominant arm
  Other Names: Meningococcal group B Vaccine
  Arms: Bexsero Group
Drug: Placebo — 2 doses administered intramuscularly at Day 0 and Day 30 in the deltoid region of the non-dominant arm
  Arms: Placebo Group

SUMMARY:
The purpose of this first time in human (FTiH) study is to assess the safety, reactogenicity and immunogenicity of 2 doses of the RSV investigational vaccine, when administered intramuscularly according to a 0, 1 month schedule, in healthy adults aged 18 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject prior to performing any study specific procedure
* A male or female between, and including, 18 and 45 years of age at the time of first vaccination
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Female subjects of non-childbearing potential may be enrolled in the study
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccina-tion, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines, or planned use during the study period
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to study vaccination, or planned administration during the study period
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine administration, with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before the first dose and ≥ 15 days after the last dose of study vaccine
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccines or planned administration during the study period
* Blood donation within 4 months prior to study entry or planned blood donation at any time during the study
* Previous vaccination against RSV
* Previous vaccination with a recombinant simian or human adenoviral vaccine
* Previous Bexsero or other vaccination against Neisseria meningitidis serogroup B
* History of or current autoimmune disease
* Family history of congenital or hereditary immunodefi-ciency
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* History of any neurological disorders or seizures
* History of transient thrombocytopenia or neurological complications following any prior vaccination
* Hypersensitivity to latex
* Hypersensitivity to Bexsero's active substances or to any of its excipients
* Allergic reaction to kanamycin
* Any medical condition that in the judgment of the investi-gator would make intramuscular injection unsafe
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Acute disease and/or fever at the time of enrolment
* Acute or chronic, clinically significant pulmonary, cardio-vascular, hepatic or renal functional abnormality, as de-termined by physical examination or laboratory screening tests
* Malignancy within previous 5 years or lymphoproliferative disorders
* Any clinically significant or any ≥ Grade 2 haematological laboratory abnormality
* Body mass index > 40 kg/m2
* Current alcohol and/or drug abuse
* Pregnant or lactating female
* Any other condition that the investigator judges may interfere with study procedures or findings
* Planned move to a location that will prohibit participating in the trial until study end

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Cicconi P, Jones C, Sarkar E, Silva-Reyes L, Klenerman P, de Lara C, Hutchings C, Moris P, Janssens M, Fissette LA, Picciolato M, Leach A, Gonzalez-Lopez A, Dieussaert I, Snape MD. First-in-Human Randomized Study to Assess the Safety and Immunogenicity of an Investigational Respiratory Syncytial Virus (RSV) Vaccine Based on Chimpanzee-Adenovirus-155 Viral Vector-Expressing RSV Fusion, Nucleocapsid, and Antitermination Viral Proteins in Healthy Adults. Clin Infect Dis. 2020 May 6;70(10):2073-2081. doi: 10.1093/cid/ciz653. PMID 31340042

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 73 subjects originally enrolled in this study, only 72 subjects received the study vaccination and were hence included in the Total Vaccinated Cohort.
Groups:
- GSK3389245A_LD Group: Subjects received 2 doses of the investigational GSK3389245A low dose (LD) vaccine, one month apart, at Day 0 and Day 30.
- GSK3389245A_HD Group: Subjects received 2 doses of the investigational GSK3389245A high dose (HD) vaccine, one month apart, at Day 0 and Day 30.
- Placebo Group: Subjects received 2 doses of placebo vaccine, one month apart, at Day 0 and Day 30.
- Bexsero Group: Subjects received 2 doses of the active control vaccine, one month apart, at Day 0 and Day 30.
Period: Overall Study
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Started | 7 | 31 | 19 | 15
Completed | 5 | 21 | 15 | 14
Not Completed | 2 | 10 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Migrated/moved from study area | 1 | 5 | 1 | 1
Not completed — Lost to Follow-up | 0 | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group | Total
Number analyzed (Participants) | 7 | 31 | 19 | 15 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.9 (8.2) | 30.6 (8.7) | 31.3 (8.6) | 29.5 (7.6) | 30.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 12 | 10 | 41
  Male | 2 | 17 | 7 | 5 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - Central/South Asian Heritage | 0 | 3 | 1 | 0 | 4
  Geographic ancestry: Asian - East Asian Heritage | 0 | 1 | 0 | 0 | 1
  Geographic ancestry: Asian - Japanese Heritage | 0 | 0 | 1 | 0 | 1
  Geographic ancestry: Asian - South East Asian Heritage | 0 | 1 | 0 | 0 | 1
  Geographic ancestry: White - Caucasian / European Heritage | 7 | 26 | 17 | 14 | 64
  Geographic ancestry: Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. All solicited local symptoms are considered as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administration documented, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 30 | 19 | 15
Participants
  Any Pain Dose 1 | 2 | 23 | 1 | 15
  Grade 3 Pain Dose 1 | 0 | 1 | 0 | 3
  Any Redness Dose 1 | 0 | 0 | 0 | 0
  Grade 3 Redness Dose 1 | 0 | 0 | 0 | 0
  Any Swelling Dose 1 | 0 | 0 | 0 | 0
  Grade 3 Swelling Dose 1 | 0 | 0 | 0 | 0
  Any Pain Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Pain Dose 2 | 2 | 19 | 0 | 15
  Grade 3 Pain Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Pain Dose 2 | 0 | 1 | 0 | 2
  Any Redness Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Redness Dose 2 | 0 | 0 | 0 | 3
  Grade 3 Redness Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Redness Dose 2 | 0 | 0 | 0 | 1
  Any Swelling Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Swelling Dose 2 | 0 | 0 | 0 | 1
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Swelling Dose 2 | 0 | 0 | 0 | 0
  Any Pain Across doses | 4 | 27 | 1 | 15
  Grade 3 Pain Across doses | 0 | 2 | 0 | 4
  Any Redness Across doses | 0 | 0 | 0 | 3
  Grade 3 Redness Across doses | 0 | 0 | 0 | 1
  Any Swelling Across doses | 0 | 0 | 0 | 1
  Grade 3 Swelling Across doses | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)] gastrointestinal symptoms (gastro) [nausea, vomiting, diarrhoea and/or abdominal pain] and headache. Any = occurrence of the symptom regardless of intensity grade and relationship to the vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented, who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 30 | 19 | 15
Participants
  Any Fatigue Dose 1 | 3 | 19 | 8 | 8
  Grade 3 Fatigue Dose 1 | 0 | 0 | 0 | 0
  Related Fatigue Dose 1 | 3 | 19 | 8 | 8
  Any Gastro Dose 1 | 2 | 5 | 6 | 3
  Grade 3 Gastro Dose 1 | 0 | 0 | 0 | 0
  Related Gastro Dose 1 | 2 | 5 | 6 | 3
  Any Headache Dose 1 | 5 | 14 | 8 | 10
  Grade 3 Headache Dose 1 | 1 | 0 | 0 | 0
  Related Headache Dose 1 | 5 | 14 | 8 | 10
  Any Fever Dose 1 | 0 | 5 | 0 | 1
  Grade 3 Fever Dose 1 | 0 | 0 | 0 | 0
  Related Fever Dose 1 | 0 | 5 | 0 | 1
  Any Fatigue Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Fatigue Dose 2 | 1 | 10 | 6 | 9
  Grade 3 Fatigue Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Fatigue Dose 2 | 0 | 1 | 0 | 0
  Related Fatigue Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Related Fatigue Dose 2 | 1 | 10 | 6 | 9
  Any Gastro Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Gastro Dose 2 | 2 | 4 | 4 | 2
  Grade 3 Gastro Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Gastro Dose 2 | 0 | 0 | 0 | 0
  Related Gastro Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Related Gastro Dose 2 | 1 | 4 | 4 | 1
  Any Headache Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Headache Dose 2 | 1 | 6 | 5 | 9
  Grade 3 Headache Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Headache Dose 2 | 0 | 0 | 0 | 0
  Related Headache Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Related Headache Dose 2 | 1 | 6 | 5 | 9
  Any Fever Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Any Fever Dose 2 | 0 | 4 | 1 | 2
  Grade 3 Fever Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Grade 3 Fever Dose 2 | 0 | 0 | 0 | 0
  Related Fever Dose 2: number analyzed (Participants) | 7 | 28 | 19 | 15
  Related Fever Dose 2 | 0 | 4 | 1 | 2
  Any Fatigue Across doses | 4 | 19 | 9 | 11
  Grade 3 Fatigue Across doses | 0 | 1 | 0 | 0
  Related Fatigue Across doses | 4 | 19 | 9 | 11
  Any Gastro Across doses | 3 | 7 | 9 | 4
  Grade 3 Gastro Across doses | 0 | 0 | 0 | 0
  Related Gastro Across doses | 2 | 7 | 9 | 4
  Any Headache Across doses | 5 | 16 | 10 | 12
  Grade 3 Headache Across doses | 1 | 0 | 0 | 0
  Related Headache Across doses | 5 | 16 | 10 | 12
  Any Fever Across doses | 0 | 8 | 1 | 2
  Grade 3 Fever Across doses | 0 | 0 | 0 | 0
  Related Fever Across doses | 0 | 8 | 1 | 2

3. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cells [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 1 (U-B), unknown at baseline and within at Day 1 (U-W), unknown at baseline and above at Day 1 (U-A), below at baseline and below at Day 1 (B-B), below at baseline and within at Day 1 (B-W), below at baseline and above at Day 1(B-A), within at baseline and below at Day 1 (W-B), within at baseline and within at Day 1(W-W), within at baseline and above at Day 1(W-A), above at baseline and below at Day 1(A-B), above at baseline and within at Day 1 (A-W), above at baseline and above at Day 1(A-A)
Time Frame: At Day 1
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 31 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-W | 7 | 29 | 18 | 11
  PTT, W-A: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-A | 0 | 0 | 0 | 1
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 1
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 2 | 1 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 0 | 0 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-B | 0 | 0 | 2 | 2
  ALT, W-W: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-W | 7 | 27 | 13 | 12
  ALT, W-A: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-A | 0 | 0 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 2 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 2 | 3 | 1
  ALT, A-W | 0 | 0 | 1 | 0
  ALT, A-A: number analyzed (Participants) | 0 | 2 | 3 | 1
  ALT, A-A | 0 | 2 | 2 | 1
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, W-B | 1 | 0 | 0 | 0
  AST, W-W: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, W-W | 6 | 29 | 19 | 15
  AST, W-A: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, W-A | 0 | 1 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-W | 5 | 22 | 13 | 9
  BLD, W-A: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-A | 1 | 5 | 3 | 5
  BLD, A-B: number analyzed (Participants) | 1 | 4 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 4 | 3 | 1
  BLD, A-W | 0 | 0 | 1 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 4 | 3 | 1
  BLD, A-A | 1 | 4 | 2 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-B | 0 | 1 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-W | 7 | 24 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-A | 0 | 0 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 4 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 4 | 0 | 0
  CRE, A-W | 0 | 2 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 4 | 0 | 0
  CRE, A-A | 0 | 2 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 30 | 19 | 13
  EOS, W-B | 0 | 3 | 0 | 1
  EOS, W-W: number analyzed (Participants) | 6 | 30 | 19 | 13
  EOS, W-W | 6 | 27 | 18 | 12
  EOS, W-A: number analyzed (Participants) | 6 | 30 | 19 | 13
  EOS, W-A | 0 | 0 | 1 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 0
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 1
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-B | 0 | 2 | 0 | 1
  RBC, W-W: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-W | 6 | 24 | 11 | 13
  RBC, W-A: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-A | 1 | 0 | 1 | 1
  RBC, A-B: number analyzed (Participants) | 0 | 5 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 5 | 7 | 0
  RBC, A-W | 0 | 0 | 4 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 5 | 7 | 0
  RBC, A-A | 0 | 5 | 3 | 0
  Hpg, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  Hpg, B-B | 1 | 1 | 2 | 0
  Hpg, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  Hpg, B-W | 0 | 2 | 0 | 1
  Hpg, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  Hpg, B-A | 0 | 0 | 0 | 0
  Hpg, W-B: number analyzed (Participants) | 6 | 27 | 17 | 14
  Hpg, W-B | 0 | 0 | 0 | 0
  Hpg, W-W: number analyzed (Participants) | 6 | 27 | 17 | 14
  Hpg, W-W | 6 | 27 | 17 | 14
  Hpg, W-A: number analyzed (Participants) | 6 | 27 | 17 | 14
  Hpg, W-A | 0 | 0 | 0 | 0
  Hpg, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-B | 0 | 0 | 0 | 0
  Hpg, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-W | 0 | 0 | 0 | 0
  Hpg, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-A | 0 | 1 | 0 | 0
  HgL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HgL, B-B | 0 | 2 | 0 | 0
  HgL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HgL, B-W | 0 | 0 | 0 | 0
  HgL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HgL, B-A | 0 | 0 | 0 | 0
  HgL, W-B: number analyzed (Participants) | 7 | 28 | 18 | 14
  HgL, W-B | 1 | 0 | 0 | 2
  HgL, W-W: number analyzed (Participants) | 7 | 28 | 18 | 14
  HgL, W-W | 6 | 28 | 18 | 12
  HgL, W-A: number analyzed (Participants) | 7 | 28 | 18 | 14
  HgL, W-A | 0 | 0 | 0 | 0
  HgL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HgL, A-B | 0 | 0 | 0 | 0
  HgL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HgL, A-W | 0 | 0 | 1 | 1
  HgL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HgL, A-A | 0 | 1 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 23 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 23 | 16 | 12
  LDH, W-W | 5 | 22 | 16 | 12
  LDH, W-A: number analyzed (Participants) | 5 | 23 | 16 | 12
  LDH, W-A | 0 | 1 | 0 | 0
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 1 | 6 | 3 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 1 | 2 | 0 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 1 | 0 | 0 | 0
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 0 | 1 | 1 | 1
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 30 | 18 | 14
  WBC, W-B | 0 | 1 | 0 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 30 | 18 | 14
  WBC, W-W | 6 | 29 | 18 | 12
  WBC, W-A: number analyzed (Participants) | 6 | 30 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 2
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  LYM, W-B | 0 | 8 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  LYM, W-W | 7 | 21 | 19 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  LYM, W-A | 0 | 0 | 0 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 1 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 0 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, W-B | 0 | 1 | 1 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, W-W | 6 | 30 | 17 | 11
  NEU, W-A: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, W-A | 0 | 0 | 0 | 3
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 31 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 1
  PLC, W-W: number analyzed (Participants) | 7 | 31 | 18 | 15
  PLC, W-W | 7 | 31 | 16 | 14
  PLC, W-A: number analyzed (Participants) | 7 | 31 | 18 | 15
  PLC, W-A | 0 | 0 | 2 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-W | 7 | 26 | 19 | 13
  PT, W-A: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-A | 0 | 1 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 0 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 2 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 31 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 31 | 18 | 15
  RET, W-W | 7 | 31 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 31 | 18 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-W | 7 | 27 | 19 | 14
  BLT, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-A | 0 | 2 | 0 | 1
  BLT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  BLT, A-W | 0 | 0 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  BLT, A-A | 0 | 2 | 0 | 0

4. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/ Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 3 (U-B), unknown at baseline and within at Day 3 (U-W), unknown at baseline and above at Day 3 (U-A), below at baseline and below at Day 3 (B-B), below at baseline and within at Day 3 (B-W), below at baseline and above at Day 3(B-A), within at baseline and below at Day 3 (W-B), within at baseline and within at Day 3(W-W), within at baseline and above at Day 3(W-A), above at baseline and below at Day 3(A-B), above at baseline and within at Day 3(A-W), above at baseline and above at Day 3(A-A).
Time Frame: At Day 3
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 3.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 30 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-W | 7 | 29 | 18 | 11
  PTT, W-A: number analyzed (Participants) | 7 | 29 | 18 | 12
  PTT, W-A | 0 | 0 | 0 | 1
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 0 | 0
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 1 | 2
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 1 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 1 | 1 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-B | 0 | 0 | 2 | 2
  ALT, W-W: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-W | 7 | 26 | 13 | 12
  ALT, W-A: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-A | 0 | 1 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 1 | 2 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 0 | 1 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-B | 1 | 0 | 0 | 0
  AST, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-W | 6 | 29 | 19 | 15
  AST, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-A | 0 | 0 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-W | 6 | 27 | 15 | 12
  BLD, W-A: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-A | 0 | 0 | 1 | 2
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 1 | 0 | 0 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 0 | 3 | 3 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-B | 0 | 2 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-W | 7 | 23 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-A | 0 | 0 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 2 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 1 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-B | 0 | 0 | 0 | 1
  EOS, W-W: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-W | 6 | 28 | 18 | 12
  EOS, W-A: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-A | 0 | 1 | 1 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 0
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 1
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-B | 1 | 2 | 1 | 2
  RBC, W-W: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-W | 5 | 24 | 10 | 13
  RBC, W-A: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-A | 1 | 0 | 1 | 0
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 3 | 6 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 1 | 1 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 1 | 2 | 0
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 2 | 0 | 1
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-B | 0 | 0 | 2 | 0
  HPG, W-W: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-W | 5 | 26 | 15 | 13
  HPG, W-A: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-A | 1 | 0 | 0 | 1
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 2 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 0 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-B | 3 | 3 | 2 | 1
  HGL, W-W: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-W | 4 | 24 | 16 | 13
  HGL, W-A: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-A | 0 | 0 | 0 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 1 | 1
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-W | 4 | 20 | 13 | 10
  LDH, W-A: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-A | 1 | 2 | 3 | 2
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 2 | 8 | 2 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 0 | 0 | 1 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 1 | 1 | 0 | 1
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 0 | 0 | 1 | 0
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-B | 0 | 0 | 1 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-W | 6 | 29 | 17 | 13
  WBC, W-A: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 1
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-W | 7 | 27 | 19 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-A | 0 | 1 | 0 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 1 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 1 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 0 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-B | 1 | 5 | 2 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-W | 5 | 25 | 16 | 13
  NEU, W-A: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-A | 0 | 0 | 0 | 1
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-W | 7 | 29 | 17 | 15
  PLC, W-A: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-A | 0 | 1 | 1 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-W | 7 | 27 | 19 | 13
  PT, W-A: number analyzed (Participants) | 7 | 27 | 19 | 13
  PT, W-A | 0 | 0 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-W | 7 | 30 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-W | 7 | 28 | 17 | 15
  BLT, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-A | 0 | 1 | 2 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/ Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 7 (U-B), unknown at baseline and within at Day 7 (U-W), unknown at baseline and above at Day 7 (U-A), below at baseline and below at Day 7 (B-B), below at baseline and within at Day 7 (B-W), below at baseline and above at Day 7(B-A), within at baseline and below at Day 7 (W-B), within at baseline and within at Day 7(W-W), within at baseline and above at Day 7(W-A), above at baseline and below at Day 7(A-B), above at baseline and within at Day 7(A-W), above at baseline and above at Day 7(A-A).
Time Frame: At Day 7
Population: The analysis was performed on the Total Vaccinated cohort which which included all subjects with at least one study vaccine administration documented and with available results at Day 7.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 30 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 0 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 1 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 29 | 17 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 29 | 17 | 12
  PTT, W-W | 7 | 29 | 17 | 11
  PTT, W-A: number analyzed (Participants) | 7 | 29 | 17 | 12
  PTT, W-A | 0 | 0 | 0 | 1
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 1
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 1
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 1
  PTT, A-A | 0 | 0 | 0 | 0
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 1 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 1 | 1 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-B | 0 | 0 | 1 | 1
  ALT, W-W: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-W | 7 | 27 | 14 | 13
  ALT, W-A: number analyzed (Participants) | 7 | 27 | 15 | 14
  ALT, W-A | 0 | 0 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 1 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 0 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-B | 1 | 0 | 0 | 1
  AST, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-W | 6 | 28 | 18 | 14
  AST, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  AST, W-A | 0 | 1 | 1 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-W | 5 | 25 | 15 | 14
  BLD, W-A: number analyzed (Participants) | 6 | 27 | 16 | 14
  BLD, W-A | 1 | 2 | 1 | 0
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 1 | 0 | 0 | 1
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 0 | 3 | 3 | 0
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-B | 0 | 2 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-W | 7 | 23 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 25 | 19 | 15
  CRE, W-A | 0 | 0 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 1 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 2 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-B | 0 | 0 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-W | 6 | 29 | 18 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 29 | 19 | 13
  EOS, W-A | 0 | 0 | 1 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 0 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 1 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-B | 1 | 0 | 0 | 1
  RBC, W-W: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-W | 5 | 26 | 12 | 12
  RBC, W-A: number analyzed (Participants) | 7 | 26 | 12 | 15
  RBC, W-A | 1 | 0 | 0 | 2
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 1 | 4 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 3 | 3 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 0
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 1
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-B | 0 | 1 | 0 | 0
  HPG, W-W: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-W | 5 | 25 | 17 | 13
  HPG, W-A: number analyzed (Participants) | 6 | 26 | 17 | 14
  HPG, W-A | 1 | 0 | 0 | 1
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 2 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 0 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-B | 0 | 0 | 1 | 1
  HGL, W-W: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-W | 7 | 27 | 16 | 13
  HGL, W-A: number analyzed (Participants) | 7 | 27 | 18 | 14
  HGL, W-A | 0 | 0 | 1 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 1 | 0
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 0 | 1
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-W | 4 | 15 | 12 | 10
  LDH, W-A: number analyzed (Participants) | 5 | 22 | 16 | 12
  LDH, W-A | 1 | 7 | 4 | 2
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 2 | 4 | 2 | 0
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 0 | 4 | 1 | 3
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 1 | 1 | 1
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 0 | 0 | 0
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-B | 0 | 0 | 1 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-W | 6 | 29 | 17 | 14
  WBC, W-A: number analyzed (Participants) | 6 | 29 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-W | 0 | 28 | 18 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 28 | 19 | 15
  LYM, W-A | 0 | 0 | 1 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 1 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 1 | 0 | 1 | 1
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 0 | 0 | 0 | 0
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-B | 0 | 2 | 2 | 1
  NEU, W-W: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-W | 6 | 27 | 15 | 13
  NEU, W-A: number analyzed (Participants) | 6 | 30 | 18 | 14
  NEU, W-A | 0 | 1 | 1 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-W | 7 | 29 | 17 | 15
  PLC, W-A: number analyzed (Participants) | 7 | 30 | 18 | 15
  PLC, W-A | 0 | 1 | 1 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 27 | 18 | 12
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 27 | 18 | 12
  PT, W-W | 7 | 26 | 17 | 11
  PT, W-A: number analyzed (Participants) | 7 | 27 | 18 | 12
  PT, W-A | 0 | 1 | 1 | 1
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-W | 7 | 30 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 30 | 18 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-W | 7 | 28 | 17 | 15
  BLT, W-A: number analyzed (Participants) | 7 | 29 | 19 | 15
  BLT, W-A | 0 | 1 | 2 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 30(U-B), unknown at baseline and within at Day30(U-W), unknown at baseline and above at Day 30(U-A), below at baseline and below at Day30(B-B), below at baseline and within at Day30(B-W), below at baseline and above at Day 30(B-A), within at baseline and below at Day 30 (W-B), within at baseline and within at Day 30(W-W), within at baseline and above at Day30(W-A), above at baseline and below at Day30(A-B), above at baseline and within at Day30(A-W), above at baseline and above at Day30(A-A).
Time Frame: At Day 30
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 30.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 27 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-W | 7 | 27 | 18 | 13
  PTT, W-A: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-A | 0 | 0 | 0 | 0
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 1
  ALT, B-B: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-B | 0 | 1 | 1 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-W | 0 | 0 | 0 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-B | 0 | 0 | 2 | 2
  ALT, W-W: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-W | 7 | 25 | 13 | 12
  ALT, W-A: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-A | 0 | 1 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 0 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 1 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B | 1 | 0 | 1 | 1
  AST, W-W | 6 | 27 | 18 | 14
  AST, W-A | 0 | 0 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 0 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 1 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-W | 4 | 24 | 16 | 11
  BLD, W-A: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-A | 2 | 1 | 0 | 3
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 1 | 0 | 2 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 0 | 3 | 1 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-W | 0 | 0 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-B | 0 | 1 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-W | 7 | 21 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-A | 0 | 1 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 2 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 1 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-B | 0 | 0 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-W | 6 | 27 | 19 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-A | 0 | 0 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-W | 1 | 0 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-A | 0 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 23 | 12 | 15
  RBC, W-B | 1 | 0 | 0 | 0
  RBC, W-W: number analyzed (Participants) | 7 | 23 | 12 | 15
  RBC, W-W | 5 | 20 | 10 | 14
  RBC, W-A: number analyzed (Participants) | 7 | 23 | 12 | 15
  RBC, W-A | 1 | 3 | 2 | 1
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 2 | 5 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 2 | 2 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 1
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 0
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 24 | 17 | 14
  HPG, W-B | 0 | 3 | 1 | 1
  HPG, W-W: number analyzed (Participants) | 6 | 24 | 17 | 14
  HPG, W-W | 6 | 21 | 15 | 13
  HPG, W-A: number analyzed (Participants) | 6 | 24 | 17 | 14
  HPG, W-A | 0 | 0 | 1 | 0
  HPG, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  HPG, A-A | 0 | 0 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 1 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 1 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 24 | 18 | 14
  HGL, W-B | 0 | 0 | 1 | 0
  HGL, W-W: number analyzed (Participants) | 7 | 24 | 18 | 14
  HGL, W-W | 7 | 24 | 16 | 14
  HGL, W-A: number analyzed (Participants) | 7 | 24 | 18 | 14
  HGL, W-A | 0 | 0 | 1 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 0 | 0
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 1 | 1
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-W | 5 | 17 | 16 | 12
  LDH, W-A: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-A | 0 | 4 | 0 | 0
  LDH, A-B: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-W | 2 | 7 | 1 | 3
  LDH, A-A: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-A | 0 | 4 | 2 | 0
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 1 | 0 | 0 | 1
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 0 | 1 | 1 | 0
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 26 | 18 | 14
  WBC, W-B | 0 | 0 | 0 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 26 | 18 | 14
  WBC, W-W | 6 | 26 | 18 | 14
  WBC, W-A: number analyzed (Participants) | 6 | 26 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-W | 7 | 26 | 18 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-A | 0 | 0 | 1 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  LYM, A-A | 0 | 0 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 1 | 0 | 0 | 1
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 0 | 0 | 1 | 0
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 27 | 18 | 14
  NEU, W-B | 0 | 1 | 1 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 27 | 18 | 14
  NEU, W-W | 5 | 26 | 17 | 14
  NEU, W-A: number analyzed (Participants) | 6 | 27 | 18 | 14
  NEU, W-A | 1 | 0 | 0 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 27 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 7 | 27 | 18 | 15
  PLC, W-W | 7 | 26 | 17 | 15
  PLC, W-A: number analyzed (Participants) | 7 | 27 | 18 | 15
  PLC, W-A | 0 | 1 | 1 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 1 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 0 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-W | 7 | 25 | 19 | 14
  PT, W-A: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-A | 0 | 0 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 27 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 27 | 18 | 15
  RET, W-W | 7 | 26 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 27 | 18 | 15
  RET, W-A | 0 | 1 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W | 7 | 26 | 18 | 14
  BLT, W-A | 0 | 1 | 1 | 1
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 0 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 1 | 0 | 0

7. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 31(U-B), unknown at baseline and within at Day31(U-W), unknown at baseline and above at Day 31(U-A), below at baseline and below at Day31(B-B), below at baseline and within at Day31(B-W), below at baseline and above at Day 31(B-A), within at baseline and below at Day 31(W-B), within at baseline and within at Day 31(W-W), within at baseline and above at Day31(W-A), above at baseline and below at Day31(A-B), above at baseline and within at Day31(A-W), above at baseline and above at Day31(A-A).
Time Frame: At Day 31
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 31.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 29 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 27 | 18 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 27 | 18 | 12
  PTT, W-W | 7 | 26 | 18 | 12
  PTT, W-A: number analyzed (Participants) | 7 | 27 | 18 | 12
  PTT, W-A | 0 | 1 | 0 | 0
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 2
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 0
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 1 | 1 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 1 | 0 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-B | 0 | 0 | 0 | 3
  ALT, W-W: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-W | 7 | 26 | 15 | 11
  ALT, W-A: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-A | 0 | 0 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 0 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 1 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 28 | 19 | 15
  AST, W-B | 1 | 1 | 0 | 2
  AST, W-W: number analyzed (Participants) | 7 | 28 | 19 | 15
  AST, W-W | 6 | 27 | 19 | 13
  AST, W-A: number analyzed (Participants) | 7 | 28 | 19 | 15
  AST, W-A | 0 | 0 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 0 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 1 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 26 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 26 | 16 | 14
  BLD, W-W | 5 | 24 | 16 | 11
  BLD, W-A: number analyzed (Participants) | 6 | 26 | 16 | 14
  BLD, W-A | 1 | 2 | 0 | 3
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 0 | 0 | 2 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 1 | 3 | 1 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-B | 0 | 0 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-W | 7 | 22 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-A | 0 | 1 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 2 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 1 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 28 | 19 | 13
  EOS, W-B | 0 | 0 | 1 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 28 | 19 | 13
  EOS, W-W | 6 | 28 | 18 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 28 | 19 | 13
  EOS, W-A | 0 | 0 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 25 | 12 | 15
  RBC, W-B | 1 | 0 | 2 | 1
  RBC, W-W: number analyzed (Participants) | 7 | 25 | 12 | 15
  RBC, W-W | 5 | 25 | 9 | 14
  RBC, W-A: number analyzed (Participants) | 7 | 25 | 12 | 15
  RBC, W-A | 1 | 0 | 1 | 0
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 2 | 4 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 2 | 3 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 1
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 0
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 25 | 17 | 14
  HPG, W-B | 0 | 1 | 2 | 0
  HPG, W-W: number analyzed (Participants) | 6 | 25 | 17 | 14
  HPG, W-W | 6 | 24 | 15 | 14
  HPG, W-A: number analyzed (Participants) | 6 | 25 | 17 | 14
  HPG, W-A | 0 | 0 | 0 | 0
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 1 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 1 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 26 | 18 | 14
  HGL, W-B | 2 | 2 | 2 | 3
  HGL, W-W: number analyzed (Participants) | 7 | 26 | 18 | 14
  HGL, W-W | 5 | 24 | 16 | 11
  HGL, W-A: number analyzed (Participants) | 7 | 26 | 18 | 14
  HGL, W-A | 0 | 0 | 0 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HGL, A-W | 0 | 0 | 0 | 0
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HGL, A-A | 0 | 1 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-W | 5 | 17 | 16 | 12
  LDH, W-A: number analyzed (Participants) | 5 | 21 | 16 | 12
  LDH, W-A | 0 | 4 | 0 | 0
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 2 | 7 | 3 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 0 | 1 | 0 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 0 | 0 | 0
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 1 | 1 | 1
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 28 | 18 | 14
  WBC, W-B | 0 | 3 | 0 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 28 | 18 | 14
  WBC, W-W | 6 | 25 | 18 | 11
  WBC, W-A: number analyzed (Participants) | 6 | 28 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 3
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 27 | 19 | 15
  LYM, W-B | 0 | 3 | 1 | 1
  LYM, W-W: number analyzed (Participants) | 7 | 27 | 19 | 15
  LYM, W-W | 7 | 24 | 16 | 13
  LYM, W-A: number analyzed (Participants) | 7 | 27 | 19 | 15
  LYM, W-A | 0 | 0 | 2 | 1
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 2 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 0 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 29 | 18 | 14
  NEU, W-B | 0 | 3 | 1 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 29 | 18 | 14
  NEU, W-W | 6 | 26 | 17 | 7
  NEU, W-A: number analyzed (Participants) | 6 | 29 | 18 | 14
  NEU, W-A | 0 | 0 | 0 | 7
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 29 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 1
  PLC, W-W: number analyzed (Participants) | 7 | 29 | 18 | 15
  PLC, W-W | 7 | 29 | 15 | 14
  PLC, W-A: number analyzed (Participants) | 7 | 29 | 18 | 15
  PLC, W-A | 0 | 0 | 3 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 25 | 19 | 13
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 25 | 19 | 13
  PT, W-W | 7 | 25 | 19 | 13
  PT, W-A: number analyzed (Participants) | 7 | 25 | 19 | 13
  PT, W-A | 0 | 0 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 0
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 1
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 29 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 29 | 18 | 15
  RET, W-W | 7 | 28 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 29 | 18 | 15
  RET, W-A | 0 | 1 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 28 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 28 | 19 | 15
  BLT, W-W | 7 | 27 | 18 | 15
  BLT, W-A: number analyzed (Participants) | 7 | 28 | 19 | 15
  BLT, W-A | 0 | 1 | 1 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 33(U-B), unknown at baseline and within at Day33(U-W), unknown at baseline and above at Day 33(U-A), below at baseline and below at Day33(B-B), below at baseline and within at Day33(B-W), below at baseline and above at Day 33 (B-A), within at baseline and below at Day 33(W-B), within at baseline and within at Day 33(W-W), within at baseline and above at Day33(W-A), above at baseline and below at Day33(A-B), above at baseline and within at Day33(A-W), above at baseline and above at Day33(A-A).
Time Frame: At Day 33
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 33.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 28 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-W | 7 | 27 | 18 | 11
  PTT, W-A: number analyzed (Participants) | 7 | 27 | 18 | 13
  PTT, W-A | 0 | 0 | 0 | 2
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 1
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 1 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 1 | 1 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 25 | 14 | 14
  ALT, W-B | 0 | 0 | 0 | 1
  ALT, W-W: number analyzed (Participants) | 7 | 25 | 14 | 14
  ALT, W-W | 7 | 24 | 14 | 13
  ALT, W-A: number analyzed (Participants) | 7 | 25 | 14 | 14
  ALT, W-A | 0 | 1 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 0 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 1 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-B | 1 | 2 | 0 | 1
  AST, W-W: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-W | 6 | 25 | 19 | 14
  AST, W-A: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-A | 0 | 0 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-W | 6 | 25 | 16 | 12
  BLD, W-A: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-A | 0 | 0 | 0 | 2
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 0 | 2 | 1 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 1 | 1 | 2 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 24 | 19 | 15
  CRE, W-B | 0 | 0 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 24 | 19 | 15
  CRE, W-W | 7 | 24 | 19 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 24 | 19 | 15
  CRE, W-A | 0 | 0 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  CRE, A-W | 0 | 1 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  CRE, A-A | 0 | 1 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-B | 0 | 0 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-W | 6 | 27 | 19 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-A | 0 | 0 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-B | 2 | 2 | 2 | 2
  RBC, W-W: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-W | 5 | 22 | 10 | 12
  RBC, W-A: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-A | 0 | 0 | 0 | 1
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 3 | 4 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 1 | 3 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 0
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 1
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 5 | 24 | 17 | 13
  HPG, W-B | 0 | 2 | 1 | 0
  HPG, W-W: number analyzed (Participants) | 5 | 24 | 17 | 13
  HPG, W-W | 5 | 22 | 16 | 12
  HPG, W-A: number analyzed (Participants) | 5 | 24 | 17 | 13
  HPG, W-A | 0 | 0 | 0 | 1
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 2 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 0 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-B | 4 | 2 | 3 | 2
  HGL, W-W: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-W | 3 | 23 | 15 | 12
  HGL, W-A: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-A | 0 | 0 | 0 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 1 | 1
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-W | 5 | 14 | 14 | 12
  LDH, W-A: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-A | 0 | 6 | 2 | 0
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 1 | 8 | 3 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 1 | 0 | 0 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 1 | 0 | 0
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 0 | 1 | 1
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-B | 0 | 1 | 0 | 1
  WBC, W-W: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-W | 6 | 26 | 18 | 13
  WBC, W-A: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-B | 0 | 0 | 0 | 1
  LYM, W-W: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-W | 7 | 26 | 18 | 14
  LYM, W-A: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-A | 0 | 0 | 1 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 1 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-B | 0 | 6 | 0 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-W | 6 | 21 | 17 | 13
  NEU, W-A: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-A | 0 | 1 | 1 | 1
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 1
  PLC, W-W: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-W | 7 | 28 | 16 | 14
  PLC, W-A: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-A | 0 | 0 | 2 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-W | 7 | 25 | 19 | 14
  PT, W-A: number analyzed (Participants) | 7 | 25 | 19 | 14
  PT, W-A | 0 | 0 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-W | 7 | 28 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-W | 7 | 26 | 19 | 14
  BLT, W-A: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-A | 0 | 1 | 0 | 1
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 37(U-B), unknown at baseline and within at Day37(U-W), unknown at baseline and above at Day 37(U-A), below at baseline and below at Day37(B-B), below at baseline and within at Day37(B-W), below at baseline and above at Day 37(B-A), within at baseline and below at Day 37(W-B), within at baseline and within at Day 37(W-W), within at baseline and above at Day37(W-A), above at baseline and below at Day37(A-B), above at baseline and within at Day37(A-W), above at baseline and above at Day37(A-A).
Time Frame: At Day 37
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 37.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 29 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 7 | 27 | 16 | 11
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 7 | 27 | 16 | 11
  PTT, W-W | 7 | 27 | 16 | 10
  PTT, W-A: number analyzed (Participants) | 7 | 27 | 16 | 11
  PTT, W-A | 0 | 0 | 0 | 1
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 1
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, B-B | 0 | 1 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, B-W | 0 | 1 | 0 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-B | 0 | 0 | 1 | 1
  ALT, W-W: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-W | 7 | 23 | 14 | 13
  ALT, W-A: number analyzed (Participants) | 7 | 26 | 15 | 14
  ALT, W-A | 0 | 3 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 0 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 1 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 28 | 17 | 15
  AST, W-B | 1 | 0 | 1 | 1
  AST, W-W: number analyzed (Participants) | 7 | 28 | 17 | 15
  AST, W-W | 6 | 26 | 15 | 14
  AST, W-A: number analyzed (Participants) | 7 | 28 | 17 | 15
  AST, W-A | 0 | 2 | 1 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 26 | 15 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 26 | 15 | 14
  BLD, W-W | 5 | 25 | 14 | 14
  BLD, W-A: number analyzed (Participants) | 6 | 26 | 15 | 14
  BLD, W-A | 1 | 1 | 1 | 0
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 0 | 1 | 2 | 1
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 1 | 2 | 1 | 0
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 23 | 18 | 15
  CRE, W-B | 0 | 0 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 23 | 18 | 15
  CRE, W-W | 7 | 23 | 18 | 14
  CRE, W-A: number analyzed (Participants) | 7 | 23 | 18 | 15
  CRE, W-A | 0 | 0 | 0 | 1
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 2 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 1 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 28 | 17 | 13
  EOS, W-B | 0 | 0 | 2 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 28 | 17 | 13
  EOS, W-W | 6 | 28 | 14 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 28 | 17 | 13
  EOS, W-A | 0 | 0 | 1 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-W | 0 | 0 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 0 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 25 | 10 | 15
  RBC, W-B | 1 | 1 | 1 | 2
  RBC, W-W: number analyzed (Participants) | 7 | 25 | 10 | 15
  RBC, W-W | 5 | 24 | 8 | 12
  RBC, W-A: number analyzed (Participants) | 7 | 25 | 10 | 15
  RBC, W-A | 1 | 0 | 1 | 1
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 2 | 6 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 2 | 1 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 0
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 1
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 25 | 15 | 14
  HPG, W-B | 0 | 2 | 1 | 0
  HPG, W-W: number analyzed (Participants) | 6 | 25 | 15 | 14
  HPG, W-W | 6 | 23 | 14 | 14
  HPG, W-A: number analyzed (Participants) | 6 | 25 | 15 | 14
  HPG, W-A | 0 | 0 | 0 | 0
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 2 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 0 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 26 | 16 | 14
  HGL, W-B | 1 | 2 | 2 | 3
  HGL, W-W: number analyzed (Participants) | 7 | 26 | 16 | 14
  HGL, W-W | 5 | 24 | 14 | 11
  HGL, W-A: number analyzed (Participants) | 7 | 26 | 16 | 14
  HGL, W-A | 1 | 0 | 0 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 1 | 1
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 21 | 15 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 21 | 15 | 12
  LDH, W-W | 5 | 19 | 10 | 10
  LDH, W-A: number analyzed (Participants) | 5 | 21 | 15 | 12
  LDH, W-A | 0 | 2 | 5 | 2
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 2 | 7 | 2 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 0 | 1 | 1 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 0 | 0 | 0
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 1 | 1 | 1
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 28 | 16 | 14
  WBC, W-B | 0 | 3 | 0 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 28 | 16 | 14
  WBC, W-W | 6 | 25 | 16 | 14
  WBC, W-A: number analyzed (Participants) | 6 | 28 | 16 | 14
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 27 | 17 | 15
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 27 | 17 | 15
  LYM, W-W | 7 | 27 | 15 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 27 | 17 | 15
  LYM, W-A | 0 | 0 | 2 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 1 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 29 | 16 | 14
  NEU, W-B | 0 | 4 | 1 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 29 | 16 | 14
  NEU, W-W | 6 | 25 | 13 | 14
  NEU, W-A: number analyzed (Participants) | 6 | 29 | 16 | 14
  NEU, W-A | 0 | 0 | 2 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 29 | 16 | 15
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 7 | 29 | 16 | 15
  PLC, W-W | 7 | 28 | 14 | 15
  PLC, W-A: number analyzed (Participants) | 7 | 29 | 16 | 15
  PLC, W-A | 0 | 1 | 2 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 7 | 25 | 17 | 12
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 7 | 25 | 17 | 12
  PT, W-W | 7 | 24 | 17 | 12
  PT, W-A: number analyzed (Participants) | 7 | 25 | 17 | 12
  PT, W-A | 0 | 1 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 29 | 16 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 29 | 16 | 15
  RET, W-W | 7 | 29 | 16 | 15
  RET, W-A: number analyzed (Participants) | 7 | 29 | 16 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 28 | 17 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 28 | 17 | 15
  BLT, W-W | 7 | 27 | 16 | 15
  BLT, W-A: number analyzed (Participants) | 7 | 28 | 17 | 15
  BLT, W-A | 0 | 1 | 1 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT]. alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day 60(U-B), unknown at baseline and within at Day60(U-W), unknown at baseline and above at Day 60(U-A), below at baseline and below at Day60(B-B), below at baseline and within at Day60(B-W), below at baseline and above at Day60(B-A), within at baseline and below at Day 60(W-B), within at baseline and within at Day 60(W-W), within at baseline and above at Day60(W-A), above at baseline and below at Day60(A-B), above at baseline and within at Day60(A-W), above at baseline and above at Day60(A-A).
Time Frame: At Day 60
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one study vaccine administration documented and with available results at Day 60.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 28 | 19 | 15
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 6 | 26 | 18 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 6 | 26 | 18 | 12
  PTT, W-W | 6 | 26 | 18 | 10
  PTT, W-A: number analyzed (Participants) | 6 | 26 | 18 | 12
  PTT, W-A | 0 | 0 | 0 | 2
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 1
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 1
  ALT, B-B: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-B | 0 | 1 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-W | 0 | 1 | 1 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 2 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 7 | 25 | 15 | 14
  ALT, W-B | 0 | 0 | 2 | 0
  ALT, W-W: number analyzed (Participants) | 7 | 25 | 15 | 14
  ALT, W-W | 7 | 24 | 13 | 14
  ALT, W-A: number analyzed (Participants) | 7 | 25 | 15 | 14
  ALT, W-A | 0 | 1 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 1 | 2 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 0 | 1 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-B | 0 | 0 | 1 | 0
  AST, W-W: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-W | 7 | 27 | 17 | 15
  AST, W-A: number analyzed (Participants) | 7 | 27 | 19 | 15
  AST, W-A | 0 | 0 | 1 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 1 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-W | 5 | 25 | 15 | 13
  BLD, W-A: number analyzed (Participants) | 6 | 25 | 16 | 14
  BLD, W-A | 1 | 0 | 1 | 1
  BLD, A-B: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-W | 1 | 1 | 0 | 1
  BLD, A-A: number analyzed (Participants) | 1 | 3 | 3 | 1
  BLD, A-A | 0 | 2 | 3 | 0
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-B | 0 | 0 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-W | 7 | 23 | 18 | 15
  CRE, W-A: number analyzed (Participants) | 7 | 23 | 19 | 15
  CRE, W-A | 0 | 0 | 1 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 1 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 2 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-B | 0 | 0 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-W | 6 | 27 | 19 | 13
  EOS, W-A: number analyzed (Participants) | 6 | 27 | 19 | 13
  EOS, W-A | 0 | 0 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 1 | 1 | 0 | 1
  EOS, A-A | 1 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-B | 0 | 3 | 1 | 0
  RBC, W-W: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-W | 5 | 20 | 11 | 14
  RBC, W-A: number analyzed (Participants) | 7 | 24 | 12 | 15
  RBC, W-A | 2 | 1 | 0 | 1
  RBC, A-B: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-W | 0 | 3 | 3 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 4 | 7 | 0
  RBC, A-A | 0 | 1 | 4 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-B | 1 | 2 | 2 | 1
  HPG, B-W: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-W | 0 | 1 | 0 | 0
  HPG, B-A: number analyzed (Participants) | 1 | 3 | 2 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 6 | 23 | 17 | 14
  HPG, W-B | 0 | 1 | 1 | 1
  HPG, W-W: number analyzed (Participants) | 6 | 23 | 17 | 14
  HPG, W-W | 6 | 22 | 16 | 13
  HPG, W-A: number analyzed (Participants) | 6 | 23 | 17 | 14
  HPG, W-A | 0 | 0 | 0 | 0
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 0 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 1 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 1 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 1 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-B | 1 | 1 | 6 | 1
  HGL, W-W: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-W | 6 | 24 | 11 | 13
  HGL, W-A: number analyzed (Participants) | 7 | 25 | 18 | 14
  HGL, W-A | 0 | 0 | 1 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-W | 0 | 1 | 1 | 1
  HGL, A-A: number analyzed (Participants) | 0 | 1 | 1 | 1
  HGL, A-A | 0 | 0 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-W | 3 | 16 | 14 | 10
  LDH, W-A: number analyzed (Participants) | 5 | 20 | 16 | 12
  LDH, W-A | 2 | 4 | 2 | 2
  LDH, A-B: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-W | 1 | 6 | 3 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 8 | 3 | 3
  LDH, A-A | 1 | 2 | 0 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 1 | 0 | 1
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 0 | 1 | 0
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-B | 0 | 1 | 1 | 0
  WBC, W-W: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-W | 6 | 26 | 17 | 14
  WBC, W-A: number analyzed (Participants) | 6 | 27 | 18 | 14
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-W | 7 | 25 | 18 | 15
  LYM, W-A: number analyzed (Participants) | 7 | 26 | 19 | 15
  LYM, W-A | 0 | 1 | 1 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 0 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 2 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 1
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 0
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-B | 0 | 4 | 0 | 0
  NEU, W-W: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-W | 6 | 22 | 18 | 14
  NEU, W-A: number analyzed (Participants) | 6 | 28 | 18 | 14
  NEU, W-A | 0 | 2 | 0 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-B | 0 | 0 | 0 | 1
  PLC, W-W: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-W | 7 | 28 | 18 | 14
  PLC, W-A: number analyzed (Participants) | 7 | 28 | 18 | 15
  PLC, W-A | 0 | 0 | 0 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 6 | 24 | 19 | 13
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 6 | 24 | 19 | 13
  PT, W-W | 6 | 24 | 18 | 13
  PT, W-A: number analyzed (Participants) | 6 | 24 | 19 | 13
  PT, W-A | 0 | 0 | 1 | 0
  PT, A-B: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 2 | 0 | 1
  PT, A-A | 0 | 1 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-W | 7 | 28 | 18 | 15
  RET, W-A: number analyzed (Participants) | 7 | 28 | 18 | 15
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-W | 7 | 26 | 18 | 15
  BLT, W-A: number analyzed (Participants) | 7 | 27 | 19 | 15
  BLT, W-A | 0 | 1 | 1 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT], alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day180(U-B), unknown at baseline and within at Day180(U-W), unknown at baseline and above at Day180(U-A), below at baseline and below at Day180(B-B), below at baseline and within at Day180(B-W),below at baseline and above at Day180(B-A), within at baseline and below at Day180(W-B),within at baseline and within at Day180(W-W), within at baseline and above at Day180(W-A),above at baseline and below at Day180(A-B),above at baseline and within at Day180(A-W),above at baseline and above at Day180(A-A).
Time Frame: At Day 180
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administration documented and with available results at Day 180.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 6 | 23 | 16 | 14
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 0 | 0 | 0
  PTT,U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT,U-A | 0 | 1 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 6 | 22 | 15 | 12
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 6 | 22 | 15 | 12
  PTT, W-W | 6 | 21 | 15 | 12
  PTT, W-A: number analyzed (Participants) | 6 | 22 | 15 | 12
  PTT, W-A | 0 | 1 | 0 | 0
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 0 | 0
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 1 | 2
  ALT, B-B: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-B | 0 | 0 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-W | 0 | 1 | 1 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 6 | 21 | 12 | 13
  ALT, W-B | 0 | 0 | 1 | 0
  ALT, W-W: number analyzed (Participants) | 6 | 21 | 12 | 13
  ALT, W-W | 5 | 21 | 11 | 13
  ALT, W-A: number analyzed (Participants) | 6 | 21 | 12 | 13
  ALT, W-A | 1 | 0 | 0 | 0
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 1 | 3 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 0 | 0 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 6 | 22 | 16 | 14
  AST, W-B | 0 | 1 | 1 | 0
  AST, W-W: number analyzed (Participants) | 6 | 22 | 16 | 14
  AST, W-W | 5 | 20 | 15 | 14
  AST, W-A: number analyzed (Participants) | 6 | 22 | 16 | 14
  AST, W-A | 1 | 1 | 0 | 0
  AST, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-W | 0 | 0 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, A-A | 0 | 1 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 5 | 21 | 13 | 13
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 5 | 21 | 13 | 13
  BLD, W-W | 4 | 21 | 11 | 11
  BLD, W-A: number analyzed (Participants) | 5 | 21 | 13 | 13
  BLD, W-A | 1 | 0 | 2 | 2
  BLD, A-B: number analyzed (Participants) | 1 | 2 | 3 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 2 | 3 | 1
  BLD, A-W | 0 | 1 | 0 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 2 | 3 | 1
  BLD, A-A | 1 | 1 | 3 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-W | 0 | 0 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 6 | 19 | 16 | 13
  CRE, W-B | 0 | 0 | 1 | 0
  CRE, W-W: number analyzed (Participants) | 6 | 19 | 16 | 13
  CRE, W-W | 6 | 19 | 15 | 13
  CRE, W-A: number analyzed (Participants) | 6 | 19 | 16 | 13
  CRE, W-A | 0 | 0 | 0 | 0
  CRE, A-B: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-W | 0 | 1 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 3 | 0 | 0
  CRE, A-A | 0 | 2 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 6 | 22 | 16 | 12
  EOS, W-B | 1 | 0 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 6 | 22 | 16 | 12
  EOS, W-W | 5 | 21 | 16 | 12
  EOS, W-A: number analyzed (Participants) | 6 | 22 | 16 | 12
  EOS, W-A | 0 | 1 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-W | 0 | 0 | 0 | 0
  EOS, A-A: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-A | 0 | 1 | 0 | 1
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 6 | 20 | 10 | 14
  RBC, W-B | 0 | 1 | 0 | 1
  RBC, W-W: number analyzed (Participants) | 6 | 20 | 10 | 14
  RBC, W-W | 5 | 16 | 9 | 11
  RBC, W-A: number analyzed (Participants) | 6 | 20 | 10 | 14
  RBC, W-A | 1 | 3 | 1 | 2
  RBC, A-B: number analyzed (Participants) | 0 | 3 | 6 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 3 | 6 | 0
  RBC, A-W | 0 | 2 | 4 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 3 | 6 | 0
  RBC, A-A | 0 | 1 | 2 | 0
  Hpg, B-B: number analyzed (Participants) | 1 | 2 | 1 | 1
  Hpg, B-B | 1 | 2 | 1 | 1
  Hpg, B-W: number analyzed (Participants) | 1 | 2 | 1 | 1
  Hpg, B-W | 0 | 0 | 0 | 0
  Hpg, B-A: number analyzed (Participants) | 1 | 2 | 1 | 1
  Hpg, B-A | 0 | 0 | 0 | 0
  Hpg, W-B: number analyzed (Participants) | 4 | 20 | 15 | 12
  Hpg, W-B | 0 | 1 | 1 | 0
  Hpg, W-W: number analyzed (Participants) | 4 | 20 | 15 | 12
  Hpg, W-W | 4 | 19 | 14 | 11
  Hpg, W-A: number analyzed (Participants) | 4 | 20 | 15 | 12
  Hpg, W-A | 0 | 0 | 0 | 1
  Hpg, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-B | 0 | 0 | 0 | 0
  Hpg, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-W | 0 | 0 | 0 | 0
  Hpg, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  Hpg, A-A | 0 | 1 | 0 | 0
  HgL, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HgL, B-B | 0 | 1 | 0 | 0
  HgL, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HgL, B-W | 0 | 0 | 0 | 0
  HgL, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HgL, B-A | 0 | 0 | 0 | 0
  HgL, W-B: number analyzed (Participants) | 6 | 22 | 16 | 13
  HgL, W-B | 1 | 2 | 1 | 1
  HgL, W-W: number analyzed (Participants) | 6 | 22 | 16 | 13
  HgL, W-W | 5 | 20 | 14 | 12
  HgL, W-A: number analyzed (Participants) | 6 | 22 | 16 | 13
  HgL, W-A | 0 | 0 | 1 | 0
  HgL, A-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  HgL, A-B | 0 | 0 | 0 | 0
  HgL, A-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  HgL, A-W | 0 | 0 | 0 | 0
  HgL, A-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  HgL, A-A | 0 | 0 | 0 | 1
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH,B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH,B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 4 | 16 | 14 | 11
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 4 | 16 | 14 | 11
  LDH, W-W | 4 | 9 | 13 | 11
  LDH, W-A: number analyzed (Participants) | 4 | 16 | 14 | 11
  LDH, W-A | 0 | 7 | 1 | 0
  LDH, A-B: number analyzed (Participants) | 2 | 7 | 2 | 2
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 7 | 2 | 2
  LDH, A-W | 1 | 3 | 1 | 1
  LDH, A-A: number analyzed (Participants) | 2 | 7 | 2 | 2
  LDH, A-A | 1 | 4 | 1 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 1 | 0 | 0
  WBC, B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-W | 1 | 0 | 1 | 1
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 5 | 22 | 15 | 13
  WBC, W-B | 0 | 1 | 2 | 0
  WBC, W-W: number analyzed (Participants) | 5 | 22 | 15 | 13
  WBC, W-W | 5 | 21 | 13 | 13
  WBC, W-A: number analyzed (Participants) | 5 | 22 | 15 | 13
  WBC, W-A | 0 | 0 | 0 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 6 | 21 | 16 | 14
  LYM, W-B | 0 | 0 | 0 | 1
  LYM, W-W: number analyzed (Participants) | 6 | 21 | 16 | 14
  LYM, W-W | 6 | 21 | 14 | 11
  LYM, W-A: number analyzed (Participants) | 6 | 21 | 16 | 14
  LYM, W-A | 0 | 0 | 2 | 2
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 1 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 1 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 0 | 0
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 1 | 1
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 5 | 23 | 15 | 13
  NEU, W-B | 0 | 2 | 1 | 0
  NEU, W-W: number analyzed (Participants) | 5 | 23 | 15 | 13
  NEU, W-W | 5 | 21 | 14 | 13
  NEU, W-A: number analyzed (Participants) | 5 | 23 | 15 | 13
  NEU, W-A | 0 | 0 | 0 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 6 | 23 | 15 | 14
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 6 | 23 | 15 | 14
  PLC, W-W | 6 | 23 | 14 | 14
  PLC, W-A: number analyzed (Participants) | 6 | 23 | 15 | 14
  PLC, W-A | 0 | 0 | 1 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 6 | 21 | 16 | 13
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 6 | 21 | 16 | 13
  PT, W-W | 6 | 21 | 15 | 13
  PT, W-A: number analyzed (Participants) | 6 | 21 | 16 | 13
  PT, W-A | 0 | 0 | 1 | 0
  PT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 1
  PT, A-W | 0 | 1 | 0 | 0
  PT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 1
  PT, A-A | 0 | 0 | 0 | 1
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 6 | 23 | 15 | 14
  RET, W-B | 0 | 0 | 0 | 0
  RET, W-W: number analyzed (Participants) | 6 | 23 | 15 | 14
  RET, W-W | 6 | 23 | 15 | 14
  RET, W-A: number analyzed (Participants) | 6 | 23 | 15 | 14
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 6 | 22 | 16 | 14
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 6 | 22 | 16 | 14
  BLT, W-W | 6 | 22 | 14 | 14
  BLT, W-A: number analyzed (Participants) | 6 | 22 | 16 | 14
  BLT, W-A | 0 | 0 | 2 | 0
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Haematological and Biochemical Laboratory Abnormalities
Description: Haematological/Biochemical parameters assessed were haemoglobin level [HgL], red blood cell [RBC], white blood cell [WBC], lymphocyte [LYM], neutrophil [NEU], eosinophil [EOS], reticulocyte [RET], platelet count [PLC], haptoglobin [Hpg], prothrombin time [PT] and partial thromboplastin time [PTT], alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CRE], lactate dehydrogenase [LDH] and bilirubin direct or total [BLD/BLT].Values were: unknown at baseline and below at Day360(U-B), unknown at baseline and within at Day360(U-W), unknown at baseline and above at Day360(U-A), below at baseline and below at Day360(B-B), below at baseline and within at Day360(B-W),below at baseline and above at Day360(B-A), within at baseline and below at Day360(W-B),within at baseline and within at Day360(W-W), within at baseline and above at Day360(W-A),above at baseline and below at Day360(A-B),above at baseline and within at Day360(A-W),above at baseline and above at Day360(A-A).
Time Frame: At Day 360
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administration documented and with available results at Day 360.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 5 | 21 | 15 | 14
Participants
  PTT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-B | 0 | 0 | 0 | 0
  PTT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-W | 0 | 1 | 0 | 0
  PTT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PTT, U-A | 0 | 0 | 0 | 0
  PTT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-B | 0 | 0 | 0 | 0
  PTT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-W | 0 | 0 | 0 | 0
  PTT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PTT, B-A | 0 | 0 | 0 | 0
  PTT, W-B: number analyzed (Participants) | 5 | 20 | 13 | 11
  PTT, W-B | 0 | 0 | 0 | 0
  PTT, W-W: number analyzed (Participants) | 5 | 20 | 13 | 11
  PTT, W-W | 5 | 19 | 13 | 10
  PTT, W-A: number analyzed (Participants) | 5 | 20 | 13 | 11
  PTT, W-A | 0 | 1 | 0 | 1
  PTT, A-B: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-B | 0 | 0 | 0 | 0
  PTT, A-W: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-W | 0 | 0 | 1 | 0
  PTT, A-A: number analyzed (Participants) | 0 | 0 | 1 | 2
  PTT, A-A | 0 | 0 | 0 | 2
  ALT, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT, B-B | 0 | 0 | 0 | 0
  ALT, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT, B-W | 0 | 1 | 0 | 0
  ALT, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT, B-A | 0 | 0 | 0 | 0
  ALT, W-B: number analyzed (Participants) | 5 | 19 | 12 | 13
  ALT, W-B | 0 | 1 | 0 | 0
  ALT, W-W: number analyzed (Participants) | 5 | 19 | 12 | 13
  ALT, W-W | 5 | 17 | 12 | 12
  ALT, W-A: number analyzed (Participants) | 5 | 19 | 12 | 13
  ALT, W-A | 0 | 1 | 0 | 1
  ALT, A-B: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-B | 0 | 0 | 0 | 0
  ALT, A-W: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-W | 0 | 1 | 2 | 1
  ALT, A-A: number analyzed (Participants) | 0 | 1 | 3 | 1
  ALT, A-A | 0 | 0 | 1 | 0
  AST, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-B | 0 | 0 | 0 | 0
  AST, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-W | 0 | 0 | 0 | 0
  AST, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, B-A | 0 | 0 | 0 | 0
  AST, W-B: number analyzed (Participants) | 5 | 21 | 14 | 14
  AST, W-B | 0 | 3 | 1 | 2
  AST, W-W: number analyzed (Participants) | 5 | 21 | 14 | 14
  AST, W-W | 5 | 18 | 13 | 11
  AST, W-A: number analyzed (Participants) | 5 | 21 | 14 | 14
  AST, W-A | 0 | 0 | 0 | 1
  AST, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, A-B | 0 | 0 | 0 | 0
  AST, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, A-W | 0 | 0 | 0 | 0
  AST, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  AST, A-A | 0 | 0 | 0 | 0
  BLD, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-B | 0 | 0 | 0 | 0
  BLD, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-W | 0 | 0 | 0 | 0
  BLD, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLD, B-A | 0 | 0 | 0 | 0
  BLD, W-B: number analyzed (Participants) | 4 | 19 | 13 | 13
  BLD, W-B | 0 | 0 | 0 | 0
  BLD, W-W: number analyzed (Participants) | 4 | 19 | 13 | 13
  BLD, W-W | 3 | 17 | 12 | 12
  BLD, W-A: number analyzed (Participants) | 4 | 19 | 13 | 13
  BLD, W-A | 1 | 2 | 1 | 1
  BLD, A-B: number analyzed (Participants) | 1 | 2 | 1 | 1
  BLD, A-B | 0 | 0 | 0 | 0
  BLD, A-W: number analyzed (Participants) | 1 | 2 | 1 | 1
  BLD, A-W | 0 | 1 | 0 | 0
  BLD, A-A: number analyzed (Participants) | 1 | 2 | 1 | 1
  BLD, A-A | 1 | 1 | 1 | 1
  CRE, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-B | 0 | 0 | 0 | 0
  CRE, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-W | 0 | 1 | 0 | 0
  CRE, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, U-A | 0 | 0 | 0 | 0
  CRE, B-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-B | 0 | 0 | 0 | 0
  CRE, B-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-W | 0 | 1 | 0 | 0
  CRE, B-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, B-A | 0 | 0 | 0 | 0
  CRE, W-B: number analyzed (Participants) | 5 | 18 | 15 | 14
  CRE, W-B | 0 | 1 | 0 | 0
  CRE, W-W: number analyzed (Participants) | 5 | 18 | 15 | 14
  CRE, W-W | 5 | 17 | 15 | 13
  CRE, W-A: number analyzed (Participants) | 5 | 18 | 15 | 14
  CRE, W-A | 0 | 0 | 0 | 1
  CRE, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, A-B | 0 | 0 | 0 | 0
  CRE, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, A-W | 0 | 1 | 0 | 0
  CRE, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, A-A | 0 | 0 | 0 | 0
  EOS, B-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-B | 0 | 0 | 0 | 1
  EOS, B-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-W | 0 | 0 | 0 | 0
  EOS, B-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  EOS, B-A | 0 | 0 | 0 | 0
  EOS, W-B: number analyzed (Participants) | 5 | 20 | 15 | 12
  EOS, W-B | 0 | 1 | 0 | 0
  EOS, W-W: number analyzed (Participants) | 5 | 20 | 15 | 12
  EOS, W-W | 5 | 19 | 15 | 12
  EOS, W-A: number analyzed (Participants) | 5 | 20 | 15 | 12
  EOS, W-A | 0 | 0 | 0 | 0
  EOS, A-B: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-B | 0 | 0 | 0 | 0
  EOS, A-W: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-W | 0 | 1 | 0 | 1
  EOS, A-A: number analyzed (Participants) | 0 | 1 | 0 | 1
  EOS, A-A | 0 | 0 | 0 | 0
  RBC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-B | 0 | 0 | 0 | 0
  RBC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-W | 0 | 0 | 0 | 0
  RBC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC, B-A | 0 | 0 | 0 | 0
  RBC, W-B: number analyzed (Participants) | 5 | 18 | 8 | 14
  RBC, W-B | 0 | 0 | 0 | 0
  RBC, W-W: number analyzed (Participants) | 5 | 18 | 8 | 14
  RBC, W-W | 5 | 17 | 7 | 12
  RBC, W-A: number analyzed (Participants) | 5 | 18 | 8 | 14
  RBC, W-A | 0 | 1 | 1 | 2
  RBC, A-B: number analyzed (Participants) | 0 | 3 | 7 | 0
  RBC, A-B | 0 | 0 | 0 | 0
  RBC, A-W: number analyzed (Participants) | 0 | 3 | 7 | 0
  RBC, A-W | 0 | 1 | 3 | 0
  RBC, A-A: number analyzed (Participants) | 0 | 3 | 7 | 0
  RBC, A-A | 0 | 2 | 4 | 0
  HPG, B-B: number analyzed (Participants) | 1 | 2 | 1 | 1
  HPG, B-B | 1 | 1 | 1 | 1
  HPG, B-W: number analyzed (Participants) | 1 | 2 | 1 | 1
  HPG, B-W | 0 | 1 | 0 | 0
  HPG, B-A: number analyzed (Participants) | 1 | 2 | 1 | 1
  HPG, B-A | 0 | 0 | 0 | 0
  HPG, W-B: number analyzed (Participants) | 4 | 18 | 13 | 13
  HPG, W-B | 0 | 1 | 0 | 1
  HPG, W-W: number analyzed (Participants) | 4 | 18 | 13 | 13
  HPG, W-W | 4 | 17 | 13 | 12
  HPG, W-A: number analyzed (Participants) | 4 | 18 | 13 | 13
  HPG, W-A | 0 | 0 | 0 | 0
  HPG, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-B | 0 | 0 | 0 | 0
  HPG, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-W | 0 | 1 | 0 | 0
  HPG, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  HPG, A-A | 0 | 0 | 0 | 0
  HGL, B-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-B | 0 | 1 | 0 | 0
  HGL, B-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-W | 0 | 1 | 0 | 0
  HGL, B-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  HGL, B-A | 0 | 0 | 0 | 0
  HGL, W-B: number analyzed (Participants) | 5 | 19 | 15 | 13
  HGL, W-B | 0 | 0 | 1 | 0
  HGL, W-W: number analyzed (Participants) | 5 | 19 | 15 | 13
  HGL, W-W | 5 | 19 | 13 | 13
  HGL, W-A: number analyzed (Participants) | 5 | 19 | 15 | 13
  HGL, W-A | 0 | 0 | 1 | 0
  HGL, A-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  HGL, A-B | 0 | 0 | 0 | 0
  HGL, A-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  HGL, A-W | 0 | 0 | 0 | 1
  HGL, A-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  HGL, A-A | 0 | 0 | 0 | 0
  LDH, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-B | 0 | 0 | 0 | 0
  LDH, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-W | 0 | 0 | 0 | 0
  LDH, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDH, B-A | 0 | 0 | 0 | 0
  LDH, W-B: number analyzed (Participants) | 3 | 14 | 11 | 11
  LDH, W-B | 0 | 0 | 0 | 0
  LDH, W-W: number analyzed (Participants) | 3 | 14 | 11 | 11
  LDH, W-W | 3 | 12 | 11 | 10
  LDH, W-A: number analyzed (Participants) | 3 | 14 | 11 | 11
  LDH, W-A | 0 | 2 | 0 | 1
  LDH, A-B: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-B | 0 | 0 | 0 | 0
  LDH, A-W: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-W | 2 | 6 | 3 | 2
  LDH, A-A: number analyzed (Participants) | 2 | 7 | 3 | 3
  LDH, A-A | 0 | 1 | 0 | 1
  WBC, B-B: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-B | 0 | 1 | 1 | 1
  WBC,B-W: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC,B-W | 1 | 0 | 0 | 0
  WBC, B-A: number analyzed (Participants) | 1 | 1 | 1 | 1
  WBC, B-A | 0 | 0 | 0 | 0
  WBC, W-B: number analyzed (Participants) | 4 | 20 | 14 | 13
  WBC, W-B | 0 | 1 | 0 | 1
  WBC, W-W: number analyzed (Participants) | 4 | 20 | 14 | 13
  WBC, W-W | 4 | 18 | 13 | 12
  WBC, W-A: number analyzed (Participants) | 4 | 20 | 14 | 13
  WBC, W-A | 0 | 1 | 1 | 0
  WBC, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-B | 0 | 0 | 0 | 0
  WBC, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-W | 0 | 0 | 0 | 0
  WBC, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC, A-A | 0 | 0 | 0 | 0
  LYM, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-B | 0 | 0 | 0 | 0
  LYM, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-W | 0 | 0 | 0 | 0
  LYM, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM, B-A | 0 | 0 | 0 | 0
  LYM, W-B: number analyzed (Participants) | 5 | 19 | 15 | 14
  LYM, W-B | 0 | 0 | 0 | 0
  LYM, W-W: number analyzed (Participants) | 5 | 19 | 15 | 14
  LYM, W-W | 5 | 18 | 14 | 14
  LYM, W-A: number analyzed (Participants) | 5 | 19 | 15 | 14
  LYM, W-A | 0 | 1 | 1 | 0
  LYM, A-B: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-B | 0 | 0 | 0 | 0
  LYM, A-W: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-W | 0 | 2 | 0 | 0
  LYM, A-A: number analyzed (Participants) | 0 | 2 | 0 | 0
  LYM, A-A | 0 | 0 | 0 | 0
  NEU, B-B: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-B | 0 | 0 | 1 | 1
  NEU, B-W: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-W | 1 | 0 | 0 | 0
  NEU, B-A: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, B-A | 0 | 0 | 0 | 0
  NEU, W-B: number analyzed (Participants) | 4 | 21 | 14 | 13
  NEU, W-B | 0 | 3 | 0 | 1
  NEU, W-W: number analyzed (Participants) | 4 | 21 | 14 | 13
  NEU, W-W | 4 | 17 | 13 | 12
  NEU, W-A: number analyzed (Participants) | 4 | 21 | 14 | 13
  NEU, W-A | 0 | 1 | 1 | 0
  NEU, A-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-B | 0 | 0 | 0 | 0
  NEU, A-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-W | 0 | 0 | 0 | 0
  NEU, A-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU, A-A | 0 | 0 | 0 | 0
  PLC, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-B | 0 | 0 | 0 | 0
  PLC, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-W | 0 | 0 | 0 | 0
  PLC, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLC, B-A | 0 | 0 | 0 | 0
  PLC, W-B: number analyzed (Participants) | 5 | 21 | 14 | 14
  PLC, W-B | 0 | 0 | 0 | 0
  PLC, W-W: number analyzed (Participants) | 5 | 21 | 14 | 14
  PLC, W-W | 5 | 21 | 12 | 14
  PLC, W-A: number analyzed (Participants) | 5 | 21 | 14 | 14
  PLC, W-A | 0 | 0 | 2 | 0
  PLC, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-B | 0 | 0 | 0 | 0
  PLC, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-W | 0 | 0 | 0 | 0
  PLC, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  PLC, A-A | 0 | 0 | 1 | 0
  PT, U-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-B | 0 | 0 | 0 | 0
  PT, U-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-W | 0 | 1 | 0 | 0
  PT, U-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, U-A | 0 | 0 | 0 | 0
  PT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-B | 0 | 0 | 0 | 0
  PT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-W | 0 | 0 | 0 | 0
  PT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  PT, B-A | 0 | 0 | 0 | 0
  PT, W-B: number analyzed (Participants) | 5 | 20 | 14 | 12
  PT, W-B | 0 | 0 | 0 | 0
  PT, W-W: number analyzed (Participants) | 5 | 20 | 14 | 12
  PT, W-W | 5 | 20 | 14 | 12
  PT, W-A: number analyzed (Participants) | 5 | 20 | 14 | 12
  PT, W-A | 0 | 0 | 0 | 0
  PT, A-B: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, A-B | 0 | 0 | 0 | 0
  PT, A-W: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, A-W | 0 | 0 | 0 | 1
  PT, A-A: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, A-A | 0 | 0 | 0 | 0
  RET, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-B | 0 | 0 | 0 | 0
  RET, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-W | 0 | 0 | 0 | 0
  RET, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  RET, B-A | 0 | 0 | 0 | 0
  RET, W-B: number analyzed (Participants) | 5 | 21 | 13 | 14
  RET, W-B | 0 | 0 | 1 | 0
  RET, W-W: number analyzed (Participants) | 5 | 21 | 13 | 14
  RET, W-W | 5 | 21 | 12 | 14
  RET, W-A: number analyzed (Participants) | 5 | 21 | 13 | 14
  RET, W-A | 0 | 0 | 0 | 0
  RET, A-B: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-B | 0 | 0 | 0 | 0
  RET, A-W: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-W | 0 | 0 | 0 | 0
  RET, A-A: number analyzed (Participants) | 0 | 0 | 1 | 0
  RET, A-A | 0 | 0 | 1 | 0
  BLT, B-B: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-B | 0 | 0 | 0 | 0
  BLT, B-W: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-W | 0 | 0 | 0 | 0
  BLT, B-A: number analyzed (Participants) | 0 | 0 | 0 | 0
  BLT, B-A | 0 | 0 | 0 | 0
  BLT, W-B: number analyzed (Participants) | 5 | 20 | 15 | 14
  BLT, W-B | 0 | 0 | 0 | 0
  BLT, W-W: number analyzed (Participants) | 5 | 20 | 15 | 14
  BLT, W-W | 5 | 20 | 14 | 13
  BLT, W-A: number analyzed (Participants) | 5 | 20 | 15 | 14
  BLT, W-A | 0 | 0 | 1 | 1
  BLT, A-B: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-B | 0 | 0 | 0 | 0
  BLT, A-W: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-W | 0 | 1 | 0 | 0
  BLT, A-A: number analyzed (Participants) | 0 | 1 | 0 | 0
  BLT, A-A | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Subjects With Haematological and Biochemical Results by Maximum Grade
Description: Parameters analysed were ALT, activated partial thromboplastin time [APTT], AST, total bilirubin [TB], CRE, EOS, haemoglobin decrease [HgD], LYM, NEU, platelets [PLA], PT, white blood cells decrease [WBCD] and white blood cells increase [WBCI]. Assessed grades were: Unknown [UG], grade 0 [G0] = no grade, 1 [G1] = mild grade, 2 [G2] = moderate grade, 3 [G3] = severe grade, 4 [G4] = potentially life threatening and overall grading [GTotal]. Parameter grade combinations expressed were: parameter plus UG/G0/1/2/3/4/Total at baseline versus grading G0/1/2/3/4/Total from Day 1 up to Day 60, for the same parameter, e.g. ALT G0-G2.
Time Frame: From Day 1 to Day 60
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 31 | 19 | 15
Participants
  ALT, G0-G0: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G0 | 7 | 25 | 17 | 14
  ALT, G0-G1: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G1 | 0 | 4 | 0 | 1
  ALT, G0-G2: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G2 | 0 | 0 | 0 | 0
  ALT, G0-G3: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G3 | 0 | 0 | 0 | 0
  ALT, G0-G4: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G4 | 0 | 0 | 0 | 0
  ALT, G1-G0: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G0 | 0 | 0 | 0 | 0
  ALT, G1-G1: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G1 | 0 | 2 | 2 | 0
  ALT, G1-G2: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G2 | 0 | 0 | 0 | 0
  ALT, G1-G3: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G3 | 0 | 0 | 0 | 0
  ALT, G1-G4: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G4 | 0 | 0 | 0 | 0
  ALT, GTotal-G0 | 7 | 25 | 17 | 14
  ALT, GTotal-G1 | 0 | 6 | 2 | 1
  ALT, GTotal-G2 | 0 | 0 | 0 | 0
  ALT, GTotal-G3 | 0 | 0 | 0 | 0
  ALT, GTotal-G4 | 0 | 0 | 0 | 0
  APTT, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G0 | 0 | 0 | 0 | 0
  APTT, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G1 | 0 | 1 | 0 | 0
  APTT, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G2 | 0 | 0 | 0 | 0
  APTT, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G3 | 0 | 0 | 0 | 0
  APTT, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G4 | 0 | 0 | 0 | 0
  APTT, G0-G0: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G0 | 7 | 29 | 18 | 11
  APTT, G0-G1: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G1 | 0 | 1 | 0 | 1
  APTT, G0-G2: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G2 | 0 | 0 | 0 | 0
  APTT, G0-G3: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G3 | 0 | 0 | 0 | 0
  APTT, G0-G4: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G4 | 0 | 0 | 0 | 0
  APTT, G1-G0: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G0 | 0 | 0 | 0 | 0
  APTT, G1-G1: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G1 | 0 | 0 | 1 | 2
  APTT, G1-G2: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G2 | 0 | 0 | 0 | 0
  APTT, G1-G3: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G3 | 0 | 0 | 0 | 0
  APTT, G1-G4: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G4 | 0 | 0 | 0 | 0
  APTT, G4-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G0 | 0 | 0 | 0 | 0
  APTT, G4-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G1 | 0 | 0 | 0 | 1
  APTT, G4-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G2 | 0 | 0 | 0 | 0
  APTT, G4-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G3 | 0 | 0 | 0 | 0
  APTT, G4-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G4 | 0 | 0 | 0 | 0
  APTT, GTotal-G0 | 7 | 29 | 18 | 11
  APTT, GTotal-G1 | 0 | 2 | 1 | 4
  APTT, GTotal-G2 | 0 | 0 | 0 | 0
  APTT, GTotal-G3 | 0 | 0 | 0 | 0
  APTT, GTotal-G4 | 0 | 0 | 0 | 0
  AST, G0-G0: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G0 | 7 | 28 | 18 | 15
  AST, G0-G1: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G1 | 0 | 2 | 1 | 0
  AST, G0-G2: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G2 | 0 | 0 | 0 | 0
  AST, G0-G3: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G3 | 0 | 0 | 0 | 0
  AST, G0-G4: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G4 | 0 | 0 | 0 | 0
  AST, G1-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G0 | 0 | 0 | 0 | 0
  AST, G1-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G1 | 0 | 1 | 0 | 0
  AST, G1-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G2 | 0 | 0 | 0 | 0
  AST, G1-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G3 | 0 | 0 | 0 | 0
  AST, G1-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G4 | 0 | 0 | 0 | 0
  AST, GTotal-G0 | 7 | 28 | 18 | 15
  AST, GTotal-G1 | 0 | 3 | 1 | 0
  AST, GTotal-G2 | 0 | 0 | 0 | 0
  AST, GTotal-G3 | 0 | 0 | 0 | 0
  AST, GTotal-G4 | 0 | 0 | 0 | 0
  TB, G0-G0: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G0 | 7 | 28 | 17 | 13
  TB, G0-G1: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G1 | 0 | 0 | 2 | 2
  TB, G0-G2: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G2 | 0 | 1 | 0 | 0
  TB, G0-G3: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G3 | 0 | 0 | 0 | 0
  TB, G0-G4: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G4 | 0 | 0 | 0 | 0
  TB, G1-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G0 | 0 | 0 | 0 | 0
  TB, G1-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G1 | 0 | 1 | 0 | 0
  TB, G1-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G2 | 0 | 0 | 0 | 0
  TB, G1-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G3 | 0 | 0 | 0 | 0
  TB, G1-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G4 | 0 | 0 | 0 | 0
  TB, G3-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G0 | 0 | 0 | 0 | 0
  TB, G3-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G1 | 0 | 0 | 0 | 0
  TB, G3-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G2 | 0 | 0 | 0 | 0
  TB, G3-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G3 | 0 | 0 | 0 | 0
  TB, G3-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G4 | 0 | 1 | 0 | 0
  TB, GTotal-G0 | 7 | 28 | 17 | 13
  TB, GTotal-G1 | 0 | 1 | 2 | 2
  TB, GTotal-G2 | 0 | 1 | 0 | 0
  TB, GTotal-G3 | 0 | 0 | 0 | 0
  TB, GTotal-G4 | 0 | 1 | 0 | 0
  CRE, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G0 | 0 | 1 | 0 | 0
  CRE, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G1 | 0 | 0 | 0 | 0
  CRE, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G2 | 0 | 0 | 0 | 0
  CRE, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G3 | 0 | 0 | 0 | 0
  CRE, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G4 | 0 | 0 | 0 | 0
  CRE, G0-G0: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G0 | 7 | 30 | 19 | 15
  CRE, G0-G1: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G1 | 0 | 0 | 0 | 0
  CRE, G0-G2: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G2 | 0 | 0 | 0 | 0
  CRE, G0-G3: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G3 | 0 | 0 | 0 | 0
  CRE, G0-G4: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G4 | 0 | 0 | 0 | 0
  CRE, GTotal-G0 | 7 | 31 | 19 | 15
  CRE, GTotal-G1 | 0 | 0 | 0 | 0
  CRE, GTotal-G2 | 0 | 0 | 0 | 0
  CRE, GTotal-G3 | 0 | 0 | 0 | 0
  CRE, GTotal-G4 | 0 | 0 | 0 | 0
  EOS, G0-G0: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G0 | 6 | 31 | 17 | 15
  EOS, G0-G1: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G1 | 0 | 0 | 2 | 0
  EOS, G0-G2: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G2 | 0 | 0 | 0 | 0
  EOS, G0-G3: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G3 | 0 | 0 | 0 | 0
  EOS, G0-G4: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G4 | 0 | 0 | 0 | 0
  EOS, G1-G0: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G0 | 0 | 0 | 0 | 0
  EOS, G1-G1: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G1 | 1 | 0 | 0 | 0
  EOS, G1-G2: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G2 | 0 | 0 | 0 | 0
  EOS, G1-G3: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G3 | 0 | 0 | 0 | 0
  EOS, G1-G4: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G4 | 0 | 0 | 0 | 0
  EOS, GTotal-G0 | 6 | 31 | 17 | 15
  EOS, GTotal-G1 | 1 | 0 | 2 | 0
  EOS, GTotal-G2 | 0 | 0 | 0 | 0
  EOS, GTotal-G3 | 0 | 0 | 0 | 0
  EOS, GTotal-G4 | 0 | 0 | 0 | 0
  HgD, G0-G0: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G0 | 2 | 22 | 12 | 10
  HgD, G0-G1: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G1 | 5 | 5 | 6 | 4
  HgD, G0-G2: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G2 | 0 | 1 | 1 | 0
  HgD, G0-G3: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G3 | 0 | 0 | 0 | 0
  HgD, G0-G4: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G4 | 0 | 0 | 0 | 0
  HgD, G1-G0: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G0 | 0 | 0 | 0 | 0
  HgD, G1-G1: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G1 | 0 | 1 | 0 | 0
  HgD, G1-G2: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G2 | 0 | 2 | 0 | 1
  HgD, G1-G3: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G3 | 0 | 0 | 0 | 0
  HgD, G1-G4: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G4 | 0 | 0 | 0 | 0
  HgD, GTotal-G0 | 2 | 22 | 12 | 10
  HgD, GTotal-G1 | 5 | 6 | 6 | 4
  HgD, GTotal-G2 | 0 | 3 | 1 | 1
  HgD, GTotal-G3 | 0 | 0 | 0 | 0
  HgD, GTotal-G4 | 0 | 0 | 0 | 0
  LYM, G0-G0 | 7 | 21 | 18 | 14
  LYM, G0-G1 | 0 | 9 | 0 | 1
  LYM, G0-G2 | 0 | 1 | 1 | 0
  LYM, G0-G3 | 0 | 0 | 0 | 0
  LYM, G0-G4 | 0 | 0 | 0 | 0
  LYM, GTotal-G0 | 7 | 21 | 18 | 14
  LYM, GTotal-G1 | 0 | 9 | 0 | 1
  LYM, GTotal-G2 | 0 | 1 | 1 | 0
  LYM, GTotal-G3 | 0 | 0 | 0 | 0
  LYM, GTotal-G4 | 0 | 0 | 0 | 0
  NEU, G0-G0: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G0 | 5 | 22 | 15 | 13
  NEU, G0-G1: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G1 | 1 | 7 | 3 | 1
  NEU, G0-G2: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G2 | 0 | 2 | 0 | 0
  NEU, G0-G3: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G3 | 0 | 0 | 0 | 0
  NEU, G0-G4: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G4 | 0 | 0 | 0 | 0
  NEU, G1-G0: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G0 | 0 | 0 | 0 | 0
  NEU, G1-G1: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G1 | 1 | 0 | 1 | 0
  NEU, G1-G2: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G2 | 0 | 0 | 0 | 1
  NEU, G1-G3: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G3 | 0 | 0 | 0 | 0
  NEU, G1-G4: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G4 | 0 | 0 | 0 | 0
  NEU, GTotal-G0 | 5 | 22 | 15 | 13
  NEU, GTotal-G1 | 2 | 7 | 4 | 1
  NEU, GTotal-G2 | 0 | 2 | 0 | 1
  NEU, GTotal-G3 | 0 | 0 | 0 | 0
  NEU, GTotal-G4 | 0 | 0 | 0 | 0
  PLA, G0-G0 | 7 | 31 | 19 | 14
  PLA, G0-G1 | 0 | 0 | 0 | 0
  PLA, G0-G2 | 0 | 0 | 0 | 1
  PLA, G0-G3 | 0 | 0 | 0 | 0
  PLA, G0-G4 | 0 | 0 | 0 | 0
  PLA, GTotal-G0 | 7 | 31 | 19 | 14
  PLA, GTotal-G1 | 0 | 0 | 0 | 0
  PLA, GTotal-G2 | 0 | 0 | 0 | 1
  PLA, GTotal-G3 | 0 | 0 | 0 | 0
  PLA, GTotal-G4 | 0 | 0 | 0 | 0
  PT, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G0 | 0 | 1 | 0 | 0
  PT, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G1 | 0 | 0 | 0 | 0
  PT, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G2 | 0 | 0 | 0 | 0
  PT, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G3 | 0 | 0 | 0 | 0
  PT, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G4 | 0 | 0 | 0 | 0
  PT, G0-G0: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G0 | 7 | 26 | 17 | 13
  PT, G0-G1: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G1 | 0 | 2 | 2 | 1
  PT, G0-G2: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G2 | 0 | 0 | 0 | 0
  PT, G0-G3: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G3 | 0 | 0 | 0 | 0
  PT, G0-G4: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G4 | 0 | 0 | 0 | 0
  PT, G1-G0: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G0 | 0 | 0 | 0 | 0
  PT, G1-G1: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G1 | 0 | 2 | 0 | 0
  PT, G1-G2: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G2 | 0 | 0 | 0 | 0
  PT, G1-G3: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G3 | 0 | 0 | 0 | 0
  PT, G1-G4: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G4 | 0 | 0 | 0 | 0
  PT, G4-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G0 | 0 | 0 | 0 | 0
  PT, G4-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G1 | 0 | 0 | 0 | 1
  PT, G4-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G2 | 0 | 0 | 0 | 0
  PT, G4-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G3 | 0 | 0 | 0 | 0
  PT, G4-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G4 | 0 | 0 | 0 | 0
  PT, GTotal-G0 | 7 | 27 | 17 | 13
  PT, GTotal-G1 | 0 | 4 | 2 | 2
  PT, GTotal-G2 | 0 | 0 | 0 | 0
  PT, GTotal-G3 | 0 | 0 | 0 | 0
  PT, GTotal-G4 | 0 | 0 | 0 | 0
  WBCD, G0-G0: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G0 | 7 | 29 | 18 | 14
  WBCD, G0-G1: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G1 | 0 | 2 | 1 | 0
  WBCD, G0-G2: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G2 | 0 | 0 | 0 | 0
  WBCD, G0-G3: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G3 | 0 | 0 | 0 | 0
  WBCD, G0-G4: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G4 | 0 | 0 | 0 | 0
  WBCD, G1-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G0 | 0 | 0 | 0 | 0
  WBCD, G1-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G1 | 0 | 0 | 0 | 1
  WBCD, G1-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G2 | 0 | 0 | 0 | 0
  WBCD, G1-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G3 | 0 | 0 | 0 | 0
  WBCD, G1-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G4 | 0 | 0 | 0 | 0
  WBCD, GTotal-G0 | 7 | 29 | 18 | 14
  WBCD, GTotal-G1 | 0 | 2 | 1 | 1
  WBCD, GTotal-G2 | 0 | 0 | 0 | 0
  WBCD, GTotal-G3 | 0 | 0 | 0 | 0
  WBCD, GTotal-G4 | 0 | 0 | 0 | 0
  WBCI, G0-G0 | 7 | 30 | 19 | 11
  WBCI, G0-G1 | 0 | 1 | 0 | 2
  WBCI, G0-G2 | 0 | 0 | 0 | 2
  WBCI, G0-G3 | 0 | 0 | 0 | 0
  WBCI, G0-G4 | 0 | 0 | 0 | 0
  WBCI, GTotal-G0 | 7 | 30 | 19 | 11
  WBCI, GTotal-G1 | 0 | 1 | 0 | 2
  WBCI, GTotal-G2 | 0 | 0 | 0 | 2
  WBCI, GTotal-G3 | 0 | 0 | 0 | 0
  WBCI, GTotal-G4 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 31 | 19 | 15
Participants | 5 | 21 | 14 | 12

15. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 to Day 360
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 31 | 19 | 15
Participants
  Up to Day 60 | 0 | 0 | 0 | 0
  Up to Day 360 | 1 | 0 | 1 | 0

16. Secondary Outcome: Number of Subjects With Haematological and Biochemical Results by Maximum Grade
Description: Parameters analysed were ALT, activated partial thromboplastin time [APTT], AST, total bilirubin [TB], CRE, EOS, haemoglobin decrease [HgD], LYM, NEU, platelets [PLA], PT, white blood cells decrease [WBCD] and white blood cells increase [WBCI]. Assessed grades were: Unknown [UG], grade 0 [G0] = no grade, 1 [G1] = mild grade, 2 [G2] = moderate grade, 3 [G3] = severe grade, 4 [G4] = potentially life threatening and overall grading [GTotal]. Parameter grade combinations expressed were: parameter plus UG/G0/1/2/3/4/Total at baseline versus grading G0/1/2/3/4/Total from Day 1 up to Day 360, for the same parameter, e.g. ALT G0-G2.
Time Frame: From Day 1 up to Day 360
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 7 | 31 | 19 | 15
Participants
  ALT, G0-G0: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G0 | 6 | 25 | 17 | 13
  ALT, G0-G1: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G1 | 1 | 4 | 0 | 2
  ALT, G0-G2: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G2 | 0 | 0 | 0 | 0
  ALT, G0-G3: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G3 | 0 | 0 | 0 | 0
  ALT, G0-G4: number analyzed (Participants) | 7 | 29 | 17 | 15
  ALT, G0-G4 | 0 | 0 | 0 | 0
  ALT, G1-G0: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G0 | 0 | 0 | 0 | 0
  ALT, G1-G1: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G1 | 0 | 2 | 2 | 0
  ALT, G1-G2: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G2 | 0 | 0 | 0 | 0
  ALT, G1-G3: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G3 | 0 | 0 | 0 | 0
  ALT, G1-G4: number analyzed (Participants) | 0 | 2 | 2 | 0
  ALT, G1-G4 | 0 | 0 | 0 | 0
  ALT, GTotal-G0 | 6 | 25 | 17 | 13
  ALT, GTotal-G1 | 1 | 6 | 2 | 2
  ALT, GTotal-G2 | 0 | 0 | 0 | 0
  ALT, GTotal-G3 | 0 | 0 | 0 | 0
  ALT, GTotal-G4 | 0 | 0 | 0 | 0
  APTT, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G0 | 0 | 0 | 0 | 0
  APTT, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G1 | 0 | 1 | 0 | 0
  APTT, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G2 | 0 | 0 | 0 | 0
  APTT, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G3 | 0 | 0 | 0 | 0
  APTT, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  APTT, UG-G4 | 0 | 0 | 0 | 0
  APTT, G0-G0: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G0 | 7 | 28 | 18 | 11
  APTT, G0-G1: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G1 | 0 | 2 | 0 | 1
  APTT, G0-G2: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G2 | 0 | 0 | 0 | 0
  APTT, G0-G3: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G3 | 0 | 0 | 0 | 0
  APTT, G0-G4: number analyzed (Participants) | 7 | 30 | 18 | 12
  APTT, G0-G4 | 0 | 0 | 0 | 0
  APTT, G1-G0: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G0 | 0 | 0 | 0 | 0
  APTT, G1-G1: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G1 | 0 | 0 | 1 | 2
  APTT, G1-G2: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G2 | 0 | 0 | 0 | 0
  APTT, G1-G3: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G3 | 0 | 0 | 0 | 0
  APTT, G1-G4: number analyzed (Participants) | 0 | 0 | 1 | 2
  APTT, G1-G4 | 0 | 0 | 0 | 0
  APTT, G4-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G0 | 0 | 0 | 0 | 0
  APTT, G4-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G1 | 0 | 0 | 0 | 1
  APTT, G4-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G2 | 0 | 0 | 0 | 0
  APTT, G4-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G3 | 0 | 0 | 0 | 0
  APTT, G4-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  APTT, G4-G4 | 0 | 0 | 0 | 0
  APTT, GTotal-G0 | 7 | 28 | 18 | 11
  APTT, GTotal-G1 | 0 | 3 | 1 | 4
  APTT, GTotal-G2 | 0 | 0 | 0 | 0
  APTT, GTotal-G3 | 0 | 0 | 0 | 0
  APTT, GTotal-G4 | 0 | 0 | 0 | 0
  AST, G0-G0: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G0 | 6 | 28 | 18 | 15
  AST, G0-G1: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G1 | 1 | 2 | 1 | 0
  AST, G0-G2: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G2 | 0 | 0 | 0 | 0
  AST, G0-G3: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G3 | 0 | 0 | 0 | 0
  AST, G0-G4: number analyzed (Participants) | 7 | 30 | 19 | 15
  AST, G0-G4 | 0 | 0 | 0 | 0
  AST, G1-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G0 | 0 | 0 | 0 | 0
  AST, G1-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G1 | 0 | 1 | 0 | 0
  AST, G1-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G2 | 0 | 0 | 0 | 0
  AST, G1-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G3 | 0 | 0 | 0 | 0
  AST, G1-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST, G1-G4 | 0 | 0 | 0 | 0
  AST, GTotal-G0 | 6 | 28 | 18 | 15
  AST, GTotal-G1 | 1 | 3 | 1 | 0
  AST, GTotal-G2 | 0 | 0 | 0 | 0
  AST, GTotal-G3 | 0 | 0 | 0 | 0
  AST, GTotal-G4 | 0 | 0 | 0 | 0
  TB, G0-G0: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G0 | 7 | 28 | 17 | 13
  TB, G0-G1: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G1 | 0 | 0 | 2 | 2
  TB, G0-G2: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G2 | 0 | 1 | 0 | 0
  TB, G0-G3: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G3 | 0 | 0 | 0 | 0
  TB, G0-G4: number analyzed (Participants) | 7 | 29 | 19 | 15
  TB, G0-G4 | 0 | 0 | 0 | 0
  TB, G1-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G0 | 0 | 0 | 0 | 0
  TB, G1-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G1 | 0 | 1 | 0 | 0
  TB, G1-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G2 | 0 | 0 | 0 | 0
  TB, G1-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G3 | 0 | 0 | 0 | 0
  TB, G1-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G1-G4 | 0 | 0 | 0 | 0
  TB, G3-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G0 | 0 | 0 | 0 | 0
  TB, G3-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G1 | 0 | 0 | 0 | 0
  TB, G3-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G2 | 0 | 0 | 0 | 0
  TB, G3-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G3 | 0 | 0 | 0 | 0
  TB, G3-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  TB, G3-G4 | 0 | 1 | 0 | 0
  TB, GTotal-G0 | 7 | 28 | 17 | 13
  TB, GTotal-G1 | 0 | 1 | 2 | 2
  TB, GTotal-G2 | 0 | 1 | 0 | 0
  TB, GTotal-G3 | 0 | 0 | 0 | 0
  TB, GTotal-G4 | 0 | 1 | 0 | 0
  CRE, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G0 | 0 | 1 | 0 | 0
  CRE, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G1 | 0 | 0 | 0 | 0
  CRE, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G2 | 0 | 0 | 0 | 0
  CRE, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G3 | 0 | 0 | 0 | 0
  CRE, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  CRE, UG-G4 | 0 | 0 | 0 | 0
  CRE, G0-G0: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G0 | 7 | 30 | 19 | 15
  CRE, G0-G1: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G1 | 0 | 0 | 0 | 0
  CRE, G0-G2: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G2 | 0 | 0 | 0 | 0
  CRE, G0-G3: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G3 | 0 | 0 | 0 | 0
  CRE, G0-G4: number analyzed (Participants) | 7 | 30 | 19 | 15
  CRE, G0-G4 | 0 | 0 | 0 | 0
  CRE, GTotal-G0 | 7 | 31 | 19 | 15
  CRE, GTotal-G1 | 0 | 0 | 0 | 0
  CRE, GTotal-G2 | 0 | 0 | 0 | 0
  CRE, GTotal-G3 | 0 | 0 | 0 | 0
  CRE, GTotal-G4 | 0 | 0 | 0 | 0
  EOS, G0-G0: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G0 | 6 | 31 | 17 | 14
  EOS, G0-G1: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G1 | 0 | 0 | 2 | 1
  EOS, G0-G2: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G2 | 0 | 0 | 0 | 0
  EOS, G0-G3: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G3 | 0 | 0 | 0 | 0
  EOS, G0-G4: number analyzed (Participants) | 6 | 31 | 19 | 15
  EOS, G0-G4 | 0 | 0 | 0 | 0
  EOS, G1-G0: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G0 | 0 | 0 | 0 | 0
  EOS, G1-G1: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G1 | 1 | 0 | 0 | 0
  EOS, G1-G2: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G2 | 0 | 0 | 0 | 0
  EOS, G1-G3: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G3 | 0 | 0 | 0 | 0
  EOS, G1-G4: number analyzed (Participants) | 1 | 0 | 0 | 0
  EOS, G1-G4 | 0 | 0 | 0 | 0
  EOS, GTotal-G0 | 6 | 31 | 17 | 14
  EOS, GTotal-G1 | 1 | 0 | 2 | 1
  EOS, GTotal-G2 | 0 | 0 | 0 | 0
  EOS, GTotal-G3 | 0 | 0 | 0 | 0
  EOS, GTotal-G4 | 0 | 0 | 0 | 0
  HgD, G0-G0: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G0 | 2 | 22 | 12 | 9
  HgD, G0-G1: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G1 | 5 | 4 | 5 | 5
  HgD, G0-G2: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G2 | 0 | 2 | 2 | 0
  HgD, G0-G3: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G3 | 0 | 0 | 0 | 0
  HgD, G0-G4: number analyzed (Participants) | 7 | 28 | 19 | 14
  HgD, G0-G4 | 0 | 0 | 0 | 0
  HgD, G1-G0: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G0 | 0 | 0 | 0 | 0
  HgD, G1-G1: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G1 | 0 | 1 | 0 | 0
  HgD, G1-G2: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G2 | 0 | 2 | 0 | 1
  HgD, G1-G3: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G3 | 0 | 0 | 0 | 0
  HgD, G1-G4: number analyzed (Participants) | 0 | 3 | 0 | 1
  HgD, G1-G4 | 0 | 0 | 0 | 0
  HgD, GTotal-G0 | 2 | 22 | 12 | 9
  HgD, GTotal-G1 | 5 | 5 | 5 | 5
  HgD, GTotal-G2 | 0 | 4 | 2 | 1
  HgD, GTotal-G3 | 0 | 0 | 0 | 0
  HgD, GTotal-G4 | 0 | 0 | 0 | 0
  LYM, G0-G0 | 7 | 21 | 18 | 13
  LYM, G0-G1 | 0 | 9 | 0 | 2
  LYM, G0-G2 | 0 | 1 | 1 | 0
  LYM, G0-G3 | 0 | 0 | 0 | 0
  LYM, G0-G4 | 0 | 0 | 0 | 0
  LYM, GTotal-G0 | 7 | 21 | 18 | 13
  LYM, GTotal-G1 | 0 | 9 | 0 | 2
  LYM, GTotal-G2 | 0 | 1 | 1 | 0
  LYM, GTotal-G3 | 0 | 0 | 0 | 0
  LYM, GTotal-G4 | 0 | 0 | 0 | 0
  NEU, G0-G0: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G0 | 5 | 21 | 14 | 13
  NEU, G0-G1: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G1 | 1 | 8 | 4 | 1
  NEU, G0-G2: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G2 | 0 | 2 | 0 | 0
  NEU, G0-G3: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G3 | 0 | 0 | 0 | 0
  NEU, G0-G4: number analyzed (Participants) | 6 | 31 | 18 | 14
  NEU, G0-G4 | 0 | 0 | 0 | 0
  NEU, G1-G0: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G0 | 0 | 0 | 0 | 0
  NEU, G1-G1: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G1 | 1 | 0 | 1 | 0
  NEU, G1-G2: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G2 | 0 | 0 | 0 | 1
  NEU, G1-G3: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G3 | 0 | 0 | 0 | 0
  NEU, G1-G4: number analyzed (Participants) | 1 | 0 | 1 | 1
  NEU, G1-G4 | 0 | 0 | 0 | 0
  NEU, GTotal-G0 | 5 | 21 | 14 | 13
  NEU, GTotal-G1 | 2 | 8 | 5 | 1
  NEU, GTotal-G2 | 0 | 2 | 0 | 1
  NEU, GTotal-G3 | 0 | 0 | 0 | 0
  NEU, GTotal-G4 | 0 | 0 | 0 | 0
  PLA, G0-G0 | 7 | 31 | 19 | 14
  PLA, G0-G1 | 0 | 0 | 0 | 0
  PLA, G0-G2 | 0 | 0 | 0 | 1
  PLA, G0-G3 | 0 | 0 | 0 | 0
  PLA, G0-G4 | 0 | 0 | 0 | 0
  PLA, GTotal-G0 | 7 | 31 | 19 | 14
  PLA, GTotal-G1 | 0 | 0 | 0 | 0
  PLA, GTotal-G2 | 0 | 0 | 0 | 1
  PLA, GTotal-G3 | 0 | 0 | 0 | 0
  PLA, GTotal-G4 | 0 | 0 | 0 | 0
  PT, UG-G0: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G0 | 0 | 1 | 0 | 0
  PT, UG-G1: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G1 | 0 | 0 | 0 | 0
  PT, UG-G2: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G2 | 0 | 0 | 0 | 0
  PT, UG-G3: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G3 | 0 | 0 | 0 | 0
  PT, UG-G4: number analyzed (Participants) | 0 | 1 | 0 | 0
  PT, UG-G4 | 0 | 0 | 0 | 0
  PT, G0-G0: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G0 | 6 | 24 | 17 | 12
  PT, G0-G1: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G1 | 1 | 4 | 2 | 2
  PT, G0-G2: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G2 | 0 | 0 | 0 | 0
  PT, G0-G3: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G3 | 0 | 0 | 0 | 0
  PT, G0-G4: number analyzed (Participants) | 7 | 28 | 19 | 14
  PT, G0-G4 | 0 | 0 | 0 | 0
  PT, G1-G0: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G0 | 0 | 0 | 0 | 0
  PT, G1-G1: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G1 | 0 | 2 | 0 | 0
  PT, G1-G2: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G2 | 0 | 0 | 0 | 0
  PT, G1-G3: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G3 | 0 | 0 | 0 | 0
  PT, G1-G4: number analyzed (Participants) | 0 | 2 | 0 | 0
  PT, G1-G4 | 0 | 0 | 0 | 0
  PT, G4-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G0 | 0 | 0 | 0 | 0
  PT, G4-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G1 | 0 | 0 | 0 | 1
  PT, G4-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G2 | 0 | 0 | 0 | 0
  PT, G4-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G3 | 0 | 0 | 0 | 0
  PT, G4-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  PT, G4-G4 | 0 | 0 | 0 | 0
  PT, GTotal-G0 | 6 | 25 | 17 | 12
  PT, GTotal-G1 | 1 | 6 | 2 | 3
  PT, GTotal-G2 | 0 | 0 | 0 | 0
  PT, GTotal-G3 | 0 | 0 | 0 | 0
  PT, GTotal-G4 | 0 | 0 | 0 | 0
  WBCD, G0-G0: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G0 | 7 | 29 | 18 | 14
  WBCD, G0-G1: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G1 | 0 | 2 | 1 | 0
  WBCD, G0-G2: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G2 | 0 | 0 | 0 | 0
  WBCD, G0-G3: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G3 | 0 | 0 | 0 | 0
  WBCD, G0-G4: number analyzed (Participants) | 7 | 31 | 19 | 14
  WBCD, G0-G4 | 0 | 0 | 0 | 0
  WBCD, G1-G0: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G0 | 0 | 0 | 0 | 0
  WBCD, G1-G1: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G1 | 0 | 0 | 0 | 1
  WBCD, G1-G2: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G2 | 0 | 0 | 0 | 0
  WBCD, G1-G3: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G3 | 0 | 0 | 0 | 0
  WBCD, G1-G4: number analyzed (Participants) | 0 | 0 | 0 | 1
  WBCD, G1-G4 | 0 | 0 | 0 | 0
  WBCD, GTotal-G0 | 7 | 29 | 18 | 14
  WBCD, GTotal-G1 | 0 | 2 | 1 | 1
  WBCD, GTotal-G2 | 0 | 0 | 0 | 0
  WBCD, GTotal-G3 | 0 | 0 | 0 | 0
  WBCD, GTotal-G4 | 0 | 0 | 0 | 0
  WBCI, G0-G0 | 7 | 29 | 18 | 11
  WBCI, G0-G1 | 0 | 2 | 1 | 2
  WBCI, G0-G2 | 0 | 0 | 0 | 2
  WBCI, G0-G3 | 0 | 0 | 0 | 0
  WBCI, G0-G4 | 0 | 0 | 0 | 0
  WBCI, GTotal-G0 | 7 | 29 | 18 | 11
  WBCI, GTotal-G1 | 0 | 2 | 1 | 2
  WBCI, GTotal-G2 | 0 | 0 | 0 | 2
  WBCI, GTotal-G3 | 0 | 0 | 0 | 0
  WBCI, GTotal-G4 | 0 | 0 | 0 | 0

17. Secondary Outcome: Anti-respiratory Syncytial Virus (RSV) Neutralizing Antibodies Titers
Description: Serum neutralizing antibody titers were reported as the inverse of the serum dilution which yielded a 60% reduction in the number of viral plaques compared to virus control without serum (Estimated Dilution: ED60). Antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: At pre-vaccination (Day 0), post-Dose 1 (Day 30) and post-Dose 2 (Day 60)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects, i.e. those who were included in the Total Vaccinated Cohort and who received at least one dose of study vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 5 | 28 | 18 | 15
Titers
  Anti-RSV, (Day 0) | 605.9 [205.1 to 1789.9] | 519.4 [349.6 to 771.7] | 346.1 [220.0 to 544.4] | 409.4 [261.8 to 640.2]
  Anti-RSV, (Day 30): number analyzed (Participants) | 5 | 26 | 18 | 15
  Anti-RSV, (Day 30) | 1474.1 [1090.0 to 1993.4] | 1293.1 [834.8 to 2002.7] | 492.4 [321.2 to 754.9] | 493.8 [318.7 to 765.3]
  Anti-RSV, (Day 60): number analyzed (Participants) | 5 | 26 | 18 | 15
  Anti-RSV, (Day 60) | 847.4 [605.6 to 1185.7] | 1211.3 [783.6 to 1872.5] | 347.3 [234.1 to 515.3] | 376.9 [220.8 to 643.3]

18. Secondary Outcome: Number of Subjects With Anti-RSV Neutralizing Antibodies Above the Cut-off Value
Description: Pre-defined cut-off values was higher than or equal to (≥) 8 ED60.
Time Frame: At pre-vaccination (Day 0), post-Dose 1 (Day 30) and post-Dose 2 (Day 60)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 5 | 28 | 18 | 15
Participants
  ANTI-RSV, (Day 0) | 5 | 28 | 18 | 15
  ANTI-RSV, (Day 30): number analyzed (Participants) | 5 | 26 | 18 | 15
  ANTI-RSV, (Day 30) | 5 | 26 | 18 | 15
  ANTI-RSV, (Day 60): number analyzed (Participants) | 5 | 26 | 18 | 15
  ANTI-RSV, (Day 60) | 5 | 26 | 18 | 15

19. Secondary Outcome: Frequency of RSV Viral Protein F, N, M2-1 Specific Interferon-gamma (IFN-γ) Secreting T-cells
Description: Interferon-gamma specific T-cells, expressed as T-cells per (/) million cells, were determined by the Enzyme Linked ImmunoSpot (ELISpot) assay.
Time Frame: At pre-vaccination (Day 0) and post-Dose 1 (Day 7, Day 30) and post-Dose 2 (Day 37, Day 60)
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 5 | 27 | 17 | 14
T-cells/million cells
  RSV F, (Day 0): number analyzed (Participants) | 5 | 26 | 16 | 14
  RSV F, (Day 0) | 33.3 [8.3 to 38.3] | 35 [13.3 to 83.3] | 15 [4.2 to 70] | 23.3 [3.3 to 38.3]
  RSV F, (Day 7): number analyzed (Participants) | 5 | 26 | 17 | 13
  RSV F, (Day 7) | 28.3 [16.7 to 33.3] | 94.2 [41.7 to 220] | 20 [3.3 to 56.7] | 36.7 [10 to 50]
  RSV F, (Day 30): number analyzed (Participants) | 5 | 27 | 15 | 12
  RSV F, (Day 30) | 1.7 [1 to 10] | 108.3 [51.7 to 175] | 41.7 [13.3 to 80] | 41.7 [6.7 to 56.7]
  RSV F, (Day 37): number analyzed (Participants) | 4 | 24 | 16 | 12
  RSV F, (Day 37) | 18 [1 to 53.3] | 75 [52.5 to 132.5] | 33.3 [7.5 to 42.5] | 35 [15 to 80]
  RSV F, (Day 60): number analyzed (Participants) | 5 | 24 | 16 | 13
  RSV F, (Day 60) | 20 [20 to 31.7] | 70.8 [35 to 155] | 52.5 [28.3 to 72.5] | 48.3 [31.7 to 80]
  RSV M2-1, (Day 0): number analyzed (Participants) | 5 | 26 | 16 | 14
  RSV M2-1, (Day 0) | 21.7 [3.3 to 31.7] | 6.7 [3.3 to 13.3] | 2.5 [1 to 8.3] | 5 [1.7 to 11.7]
  RSV M2-1, (Day 7): number analyzed (Participants) | 5 | 26 | 17 | 13
  RSV M2-1, (Day 7) | 3.3 [3.3 to 15] | 25 [1.7 to 80] | 6.7 [1.7 to 15] | 3.3 [1.7 to 15]
  RSV M2-1, (Day 30): number analyzed (Participants) | 5 | 27 | 15 | 12
  RSV M2-1, (Day 30) | 5 [1 to 13.3] | 31.7 [11.7 to 96.7] | 13.3 [1 to 41.7] | 7.5 [2.5 to 19.2]
  RSV M2-1, (Day 37): number analyzed (Participants) | 4 | 24 | 16 | 12
  RSV M2-1, (Day 37) | 20.5 [1 to 55.8] | 37.5 [21.7 to 64.2] | 5.8 [1 to 14.2] | 6.7 [2.5 to 13.3]
  RSV M2-1, (Day 60): number analyzed (Participants) | 5 | 24 | 16 | 13
  RSV M2-1, (Day 60) | 11.7 [6.7 to 11.7] | 20 [8.3 to 45.8] | 15 [6.7 to 34.5] | 10 [6.7 to 13.3]
  RSV N, (Day 0): number analyzed (Participants) | 5 | 26 | 16 | 14
  RSV N, (Day 0) | 10 [5 to 25] | 11.7 [3.3 to 25] | 5 [1 to 38.3] | 10 [1 to 25]
  RSV N, (Day 7): number analyzed (Participants) | 5 | 26 | 17 | 13
  RSV N, (Day 7) | 3.3 [1 to 30] | 21.7 [6.7 to 105] | 3.3 [1.7 to 38.3] | 11.7 [1.7 to 33.3]
  RSV N, (Day 30): number analyzed (Participants) | 5 | 27 | 15 | 12
  RSV N, (Day 30) | 1 [1 to 5] | 36.7 [21.7 to 106.7] | 18.3 [3.3 to 78.3] | 19.2 [6.7 to 31.7]
  RSV N, (Day 37): number analyzed (Participants) | 4 | 24 | 16 | 12
  RSV N, (Day 37) | 8.8 [1 to 32.5] | 50 [22.5 to 102.5] | 10.8 [3.3 to 25.8] | 18.3 [8.3 to 42.5]
  RSV N, (Day 60): number analyzed (Participants) | 5 | 24 | 16 | 13
  RSV N, (Day 60) | 15 [3.3 to 16.7] | 34.2 [15.8 to 61.7] | 24.2 [7.5 to 48.3] | 20 [10 to 73.3]

20. Secondary Outcome: Frequency of Anti-F Immunoglobulin g (IgG) and/or Immunoglobulin A (IgA) Antibody Secreting B-cells (ASC)
Description: IgG/IgA antibody specific B-cells/ expressed as B-cells per million cells, were determined by the ELISpot assay.
Time Frame: At pre-vaccination (Day 0) and post-Dose 1 (Day 7, Day 30) and post-Dose 2 (Day 37, Day 60)
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: B-cells/million cells
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
Number analyzed (Participants) | 5 | 28 | 18 | 15
B-cells/million cells
  Memory B-cell IgA, (Day 0) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgA, (Day 7): number analyzed (Participants) | 5 | 27 | 17 | 14
  Memory B-cell IgA, (Day 7) | 1 [1 to 16.7] | 16.7 [5 to 30] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgA, (Day 30): number analyzed (Participants) | 5 | 27 | 18 | 15
  Memory B-cell IgA, (Day 30) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgA, (Day 37): number analyzed (Participants) | 5 | 27 | 17 | 15
  Memory B-cell IgA, (Day 37) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgA, (Day 60): number analyzed (Participants) | 5 | 25 | 18 | 15
  Memory B-cell IgA, (Day 60) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgG, (Day 0) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgG, (Day 7): number analyzed (Participants) | 5 | 25 | 16 | 13
  Memory B-cell IgG, (Day 7) | 45 [1 to 55] | 133.3 [56.7 to 240] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgG, (Day 30): number analyzed (Participants) | 5 | 27 | 18 | 15
  Memory B-cell IgG, (Day 30) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgG, (Day 37): number analyzed (Participants) | 5 | 27 | 17 | 15
  Memory B-cell IgG, (Day 37) | 1 [1 to 1] | 1 [1 to 5] | 1 [1 to 1] | 1 [1 to 1]
  Memory B-cell IgG, (Day 60): number analyzed (Participants) | 5 | 25 | 18 | 15
  Memory B-cell IgG, (Day 60) | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited adverse events: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (up to Day 360).
Arm/Group | GSK3389245A_LD Group | GSK3389245A_HD Group | Placebo Group | Bexsero Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/31 | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/31 | 1/19 | 0/15
Other Adverse Events (participants affected / at risk) | 7/7 | 30/31 | 17/19 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3389245A_LD Group (N=7) | GSK3389245A_HD Group (N=31) | Placebo Group (N=19) | Bexsero Group (N=15)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3389245A_LD Group (N=7) | GSK3389245A_HD Group (N=31) | Placebo Group (N=19) | Bexsero Group (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (4) | 7 (9) | 9 (10) | 4 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (6) | 19 (29) | 9 (16) | 11 (17)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (4) | 27 (43) | 1 (1) | 15 (30)
Pyrexia (General disorders) | 0 (0) | 11 (13) | 1 (1) | 2 (3)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 6 (6)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sports injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (13) | 18 (35) | 11 (23) | 12 (24)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (10) | 3 (4) | 5 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.